

Av. Meridiana, 358 / 6ºplanta 08027 Barcelona Tel. 934 302 006 Fax. 934 191 768 Email: gecp@gecp.org www.gecp.org

Official Title: "A PHASE II OPEN LABEL STUDY OF ATEZOLIZUMAB IN COMBINATION WITH BEVACIZUMAB AS FIRST LINE TREATMENT FOR LOCALLY ADVANCED OR METASTASIC HIGH-INTERMEDIATE TUMOR MUTATION BURDEN (TMB) SELECTED NON-SQUAMOUS NON-SMALL CELL LUNG CANCER (NSCLC) PATIENTS" TELMA

NCT Number: NCT03836066

# **Document Dates:**

Protocol Version v.5.1 01Jul2024



Av. Meridiana, 358 / 6ªplanta 08027 Barcelona Tel. 934 302 006 Fax. 934 191 768 Email: gecp@gecp.org

www.gecp.org

# A PHASE II OPEN LABEL STUDY OF ATEZOLIZUMAB IN COMBINATION WITH BEVACIZUMAB AS FIRST LINE TREATMENT FOR LOCALLY ADVANCED OR METASTASIC HIGH-INTERMEDIATE TUMOR MUTATION BURDEN (TMB) SELECTED NON-SQUAMOUS NON-SMALL CELL LUNG CANCER (NSCLC) PATIENTS

TELMA: Atezolizumab plus bevacizumab in first line NSCLC patients

**Study Sponsor: Fundación GECP** 

EudraCT Number: 2018-004654-17

Sponsor code: GECP 18/03

Roche code:

Version 5.1



# **Contacts**

| Trial Chair | Fundación GECP<br>President | Oncology Service Hospital Univ. Puerta de Hierro, Majadahonda, Madrid, Tel. 93 430 20 06 Fax. 993 419 17 68 |
|---|---|---|
| Safety and Regulatory<br>Affairs | Coordinating office of the Fundación GECP | Avenida Meridiana 358, 6ª planta 08027 Barcelona Tel. +34 93 430 20 06 Fax. +34 93 419 17 68 |
| Coordinating office of the Fundación GECP Monitoring team | Monitor/CRA | Avenida Meridiana 358,<br>6ª planta<br>08027 Barcelona<br>Tel. +34 93 430 20 06<br>Fax. +34 93 419 17 68 |
| | Lead CRA | Avenida Meridiana 358, 6ª planta 08027 Barcelona Tel. +34 93 430 20 06 Fax. +34 93 419 17 68 |
| | Clinical Operations<br>Manager: | Avenida Meridiana 358, 6ª planta 08027 Barcelona Tel. +34 93 430 20 06 Fax. +34 93 419 17 68 |



# **Protocol Signature Page**

A PHASE II OPEN LABEL STUDY OF ATEZOLIZUMAB IN COMBINATION WITH BEVACIZUMAB AS FIRST LINE TREATMENT FOR LOCALLY ADVANCED OR METASTATIC HIGH-INTERMEDIATE TUMOR MUTATION BURDEN (TMB) SELECTED NON-SQUAMOUS NON-SMALL CELL LUNG CANCER (NSCLC) PATIENTS

TELMA: Atezolizumab plus bevacizumab in first line NSCLC patients

| Sponsor code: GECP 18/03 |
|--------------------------|
| Approved by: |
| Signature |
| Signature |
| Signature |



# **Principal Investigator Protocol Signature Page**

**Study Title:** "A phase II open-label study of Atezolizumab in combination with bevacizumab as first line treatment for locally advanced or metastatic high-intermediate tumor mutation burden (TMB) selected non-squamous non-small cell lung cancer (NSCLC) patients" **TELMA** 

Sponsor protocol code: GECP 18/03 EudraCT Number: 2018-004654-17 Protocol version: v 5.1,21th July 2024

As principal investigator of this site, I hereby confirm that:

I have read the protocol and agree that it contains all necessary details for conducting this trial. I will conduct the trial as outlined in the following protocol and in compliance with GCP and will apply due diligence to avoid protocol deviations.

I will provide copies of the protocol and all drug information relating to pre-clinical and prior clinical experience furnished to me by the Fundación GECP, to all physicians responsible to me who participate in this trial. I will discuss this material with them to assure that they are fully informed regarding the drug and the conduct of the trial.

I agree to keep accurate records on all patient information including patient's informed consent statement, drug shipment and return forms, and all other information collected during the trial for a minimum period of 25 years according to the new Royal Decree 1090/2015 approved in Spain.

| vame of Principal Investigator: | |
|---------------------------------|------|
| nstitution's name and place: | |
| Signature | Date |



# **TABLE OF CONTENTS**

| <u>Section</u> | | <u>Page</u> |
|---|---|---|
| 1. | Protocol summary | 7 |
| 2. | Trial schedule | |
| 3. | Background and rationale | 23 |
| 3.1. | Disease background and treatments in advanced NSCLC patients | 23 |
| 3.2. | Immunotherapy | 26 |
| 3.3. | Background on Atezolizumab | 26 |
| 3.4. | Background on Bevacizumab | 30 |
| 3.5. | Rationale for trial design | 31 |
| 3.6. | Rationale for additional translational research (stool and blood samples) | 32 |
| 4. | Objectives and endpoints | 33 |
| 4.1. | Primary objective and endpoint | 33 |
| 4.2. | Secondary objectives and endpoint | 34 |
| 4.3. | Exploratory objectives | 35 |
| | | 35 |
| | | 37 |
| | | 37 |
| | | 39 |
| 7. | Patient pre-screening and enrollment | 43 |
| 8. | Trial procedures | 44 |
| 8.1. | Overview of treatment sequence | 44 |
| 9. | Investigational Medicinal Product | 52 |
| 9.1. | Packaging and labelling | 53 |
| 9.2. | Receipt and storage of the IMP | 53 |
| 9.3. | Unused trial drug supplies | 53 |
| 10. | Trial treatments description | 54 |
| 10.1. | ATEZOLIZUMAB | 54 |
| 10.2. | BEVACIZUMAB | 55 |
| 11. | Dose modifications criteria | 56 |
| 11.1. | General Notes Regarding Dose Modification | 56 |
| 11.2. | ATEZOLIZUMAB dose delay criteria | 56 |
| 11.3. | BEVACIZUMAB dose delay/reduction criteria | 57 |
| 12. | Prohibited and permitted concomitant treatments | 61 |
| 13. | Adverse events and reporting | 64 |
| 13.1. | Definition of an Adverse Event (AE) and AE's reporting | 64 |
| 13.2. | Definition of Serious Adverse Event (SAE) and Suspected Unexpected Serious | Adverse |
| | Reaction (SUSAR) | |
| 13.3. | Adverse events of Special Interest for Atezolizumab (Immediately reportable | to the |
| | Sponsor) | 69 |
| | | 70 |
| 13.5. | SAEs and SUSARs reporting | 70 |
| | | 71 |
| 13.1. | Other safety considerations | 72 |
| 13.2. | Adverse events related to the treatment and associated risks | 72 |
| 14 | Riological material and translational research | 73 |



| 15. | Case report forms and documentation | 75 |
|---|---|---|
| 16. | Statistical considerations | 75 |
| 17. | Criteria for termination of the trial | 76 |
| 17.1. | General criteria for termination of the trial | 76 |
| 17.2. | Discontinuation of protocol treatment and from the study for individual patients | 77 |
| 18. | Ethics aspects, regulatory approval, and Patient Informed Consent | 78 |
| 18.1. | Ethical Review Board/Ethics Committee/Health Authority | 78 |
| 18.2. | Informed consent | |
| 19. | Governance and administrative issues | 79 |
| 19.1. | Study documentation | . 79 |
| 19.2. | Protocol non-compliances/deviations | 79 |
| 19.3. | Protocol amendment | |
| 19.4. | Final report | 80 |
| 19.5. | Independent Data Monitoring Committee | 80 |
| 19.6. | Publication | |
| 19.7. | Financial disclosure | 80 |
| 19.8. | Clinical trial insurance | 80 |
| 19.9. | Quality assurance | 80 |
| 19.10 | Data protection | 81 |
| 19.11 | . Study monitoring team | 81 |
| 19.12 | . Record retention | 82 |
| | | 82 |
| | | 86 |

# **Appendices:**

- 1. Common Terminology criteria for Adverse Events (CTCAE)
- 2. RECIST criteria v1.1
- 3. SAE Form
- 4. Pregnancy Form
- 5. Health-related Quality of life questionnaire: EORTC C30 (QLQ-C30) and submodule LC13
- 6. System of classification for non-microcytic lung cancer (NSCLC) and definition of lymph node maps, 8<sup>th</sup> edition
- 7. Risks associated with Atezolizumab and guidelines for management of adverse events associated with Atezolizumab
- 8. Patient pre-screening form TELMA
- 9. Foundation one CDx Specimen Instructions
- 10. Foundation one Liquid technical sheet
- 11. Foundation one CDx technical sheet

# **Tables:**

Table 1. Administration of First and Subsequent Infusions of Atezolizumab



# 1. Protocol summary

# A PHASE II OPEN LABEL STUDY OF ATEZOLIZUMAB IN COMBINATION WITH BEVACIZUMAB AS FIRST LINE TREATMENT FOR LOCALLY ADVANCED OR METASTATIC HIGH-INTERMEDIATE TUMOR MUTATION BURDEN (TMB) SELECTED NON-SQUAMOUS NON-SMALL CELL LUNG CANCER (NSCLC) PATIENTS

TELMA: Atezolizumab plus bevacizumab in first line NSCLC patients

**Sponsor:** Fundación GECP

Trial Chair: Mariano Provencio Pulla (MD, PhD)

Pharma Partner: Hoffmann-La Roche

Protocol code: GECP 18/03

Population: stage IIIB - IV non-squamous selected high-intermediate tumor mutation burden (TMB)

non-small cell lung cancer patients

Design: Open-label, non-randomized, phase II multi-centre clinical trial



<sup>\*</sup> If the submitted tumor sample is insufficient or not valid to evaluate the TMB, a blood sample can be sent instead .



Sample size: 40 patients

# Rationale:

Despite recent improvements in treatment, the prognosis for patients with advanced NSCLC remains dismal, with a median OS of approximately 12.5 months<sup>3</sup>.

Inhibition of programmed cell death protein-ligand 1/programmed cell death protein 1 (PD-L1/PD-1) signalling has been shown to induce durable responses in some patients with different tumors, and expression of PD-L1 by tumor cells (TCs) in several tumor types (including NSCLC) correlates with response to therapy<sup>4</sup>. Immunotherapy has demonstrated that therapies focused on enhancing T-cell responses against cancer may result in a significant survival benefit in patients with Stage IV cancer<sup>5,6,7</sup>.

Immunotherapeutic targeting of PD-L1 or PD-1 is revolutionizing the treatment of metastatic NSCLC. Currently, two anti-PD-1 therapeutic antibodies (Pembrolizumab and Nivolumab) and one anti-PD-L1 (Atezolizumab) have been approved for NSCLC treatment. Both agents are recommended as second-line agents in advanced NSCLC after prior progression on platinum-containing chemotherapy.

Atezolizumab is a humanized anti-PD-L1 monoclonal antibody that inhibits its interaction with its receptors, PD-1 and B7.1 (CD80, B7-1), reinvigorating anticancer immunity. The OAK study evaluated the efficacy of Atezolizumab compared to Docetaxel in 1.225 patients previously treated with locally-advanced or metastatic NSCLC. The PD-L1 targeted therapy by Atezolizumab resulted in a clinically relevant improvement of overall survival *versus* Docetaxel regardless of PD-L1 expression or histology, with a favourable safety profile. The median OS in this study was 13.8 months (95% CI 11.8-15.7) in the Atezolizumab arm compared to 9.6 months (95% CI 8.6-11.2) in the Docetaxel arm (HR=0.73, 95% CI 0.62-0.87; p=0.0003)<sup>8</sup>.

The GO28625 (NCT01846416, FIR) phase 2 study enrolled 137 PD-L1-selected NSCLC patients regardless previous treatments. The primary analysis for efficacy-evaluable patients, confirmed ORR after the first-line treatment with Atezolizumab was 28.6% (95% CI: 3.7-71.0) in IHC TC3 or IC3 patients and 25.8% (95% CI: 11.9-44.6) in IHC TC2/3 or IC2/3 patients<sup>9</sup>.

The efficacy and safety of Atezolizumab was also evaluated in another phase 2 single-arm study where 142 PD-L1-selected advanced NSCLC patients (NCT02031458, BIRCH) were treated with Atezolizumab monotherapy. The primary endpoint ORR in the ITT population was 25%, in TC3 or IC3 subgroup was 34% and 18% in TC2 and IC2. Median PFS and OS for the entire population were 7.3 and 23.5 months respectively. These results indicate that Atezolizumab monotherapy has durable efficacy in the first line setting<sup>10</sup>.

Currently, first-line treatment for advanced NSCLC without presence of genetic aberrations, such as sensitizing mutations of epidermal growth factor receptor (EGFR) or translocations of anaplastic lymphoma kinase (ALK), are chemotherapy and Pembrolizumab, approved based on KEYNOTE-024 study. This study randomized patients with advanced NSCLC and PD-L1 expression (at least 50% of



tumor cells), showing median progression-free survival (PFS) of 10.3 months (95% CI 6.7-not reached) versus 6.0 months (95% CI 4.2-6.2) (HR 0.50; 95% CI 0.37-0.68; P<0.001) for the Pembrolizumab and chemotherapy groups respectively<sup>11</sup>.

Currently there is a clinical trial (NCT02409342, IMpower110) of Atezolizumab as first line monotherapy in PD-L1 selected NSCLC patients that is expected to add the first line approval to Roche's portfolio. Thus, all the above data support the rational of cancer immunotherapy in first line PD-L1 positive NSCLC<sup>12</sup>. In addition, there is a growing body of evidence that suggests that proangiogenic factors can modulate the immune response and may serve as mechanisms of scape. Therefore, the combination of cancer immunotherapy with antiangiogenic agents makes sense.

The vascular endothelial growth factor (VEGF) is the most important pro-angiogenic protein and a key regulator of physiological angiogenesis. It is also implicated in pathological angiogenesis associated with tumor growth. Indeed, increased levels of VEGF have been found in lung cancer; moreover, the overexpression of VEGF is associated with a poor prognosis<sup>13,14</sup>. Actually, VEGF plays a role in cancer immune evasion through modification of the endothelial cells in the tumor microenvironment, where VEGF may reduce lymphocyte adhesion and migration from vessels to the tumor site contributing to decreased immune cell recruitment<sup>15</sup>. Given the immunosuppressive role of VEGF and angiogenesis within tumors, it is not surprising that there is evidence supporting how antiangiogenic agents stimulate the immune response and enhance the efficacy of immunotherapies<sup>16</sup>.

Recent findings indicating an intertwined regulation of VEGF signalling and immunosuppression in the tumor microenvironment suggest that the combination of anti-VEGF agents and immune checkpoint blockade could have synergistic antitumor activity, along with favourable tolerability<sup>16</sup>.

Bevacizumab is a recombinant, humanized therapeutic anti-VEGF antibody that inhibits tumor angiogenesis which may correct the immunosuppressive function exerted by VEGF, increasing the infiltration of T effector cells in cancer<sup>17</sup>.

So far, the more advanced studies to address the combination of cancer immunotherapy (CIT)-antiangiogenic agents such as Bevacizumab, there is a phase 3 study of Paclitaxel, Carboplatin Bevacizumab and Atezolizumab (NCT02366143, IMpower150). IMpower150 is the first phase III immunotherapy-based combination study to demonstrate a statistically significant and clinically meaningful improvement in PFS in all-comer 1L NSQ mNSCLC, providing a potential new standard of care for patients, showing a median PFS of 8.3 moths vs 6.8 moths (HR 0.62; 95% CI: 0.52, 0.74; P < 0.0001) for the Atezolizumab, chemotherapy and Bevacizumab arm (ABCP) and Carboplatin, Paclitaxel and Bevacizumab arm (BCP) respectively. In terms of PFS 12 months the results were 37% in the Atezolizumab arm vs 18% un the CT + Bevacizumab arm. Median overall survival among the patients was longer in the ABCP group than in the BCP group (19.2 months vs. 14.7 months; hazard ratio for death, 0.78; 95% CI, 0.64 to 0.96; P = 0.02)<sup>18</sup>.

The phase 3 study of Atezolizumab in combination with Bevacizumab compared to Sunitinib single agent (IMmotion151), as first-line therapy in untreated metastatic Renal Cell Carcinoma (RCC) patients. This clinical trial showed a significant benefit of 3.5 months in the PFS favouring the CIT-Bevacizumab combination (11.2 m vs. 7.7 m) with a tolerable safety profile in PD-L1+ patients<sup>19</sup>.



These data confirm the role of Bevacizumab as an immune modulating agent that may provide a successful combination strategy in different tumor types.

Increased mutation rate is a well-characterized feature of human cancer. Abnormal activity in several cellular pathways, including DNA damage repair and DNA replication, can increase the overall rate of somatic mutations in tumors, as can exposure to mutagens such as ultraviolet light and tobacco smoke<sup>20</sup>. Defects in DNA damage repair lead to the accumulation of mutations caused by replicative errors and environmental damage<sup>21</sup>.

The core DNA mismatch repair protein complex is composed of two cooperative dimers: the PMS2 protein dimerizes with MLH1 to form the complex MutL-alpha, which cooperates with the MSH2-MSH6 dimer, MutS-alpha, to repair single base pair mismatches and small insertion—deletion loops<sup>22</sup>. PMS2 promoter mutations are present in ~10% of melanoma samples and ~8% of squamous cell carcinomas<sup>23</sup>.

Perturbations in mismatch repair gene expression, both loss and overexpression, can be deleterious to genomic stability, and loss of function mutations in mismatch repair pathway genes are known to correlate with high Tumor Mutational Burden (TMB) in tumors, overall mutations in these genes accounted for less than 10% of cases with high TMB<sup>23</sup>.

As such, tumors with defective DNA repair mechanisms are more likely to benefit from immunotherapy. DNA replication is another key pathway in which defects can lead to increased somatic mutation rate.

Loss of function mutations in TP53 are very common in cancer and are a somatic marker of elevated mutation rate<sup>24</sup>. Mutations in a number of other genes have also been linked to increase TMB. KRASmutant lung cancers account for approximately 25% of non-small cell lung carcinomas, thus representing an enormous burden of cancer worldwide. KRAS mutations are clear drivers of tumor growth and are characterized by a complex biology involving the interaction between mutant KRAS, various growth factor pathways, and tumor suppressor genes. KRAS mutations are classically associated with a significant smoking history<sup>25</sup>. Then, it is an emerging biomarker for response to immunotherapy. The CheckMate 026 trial is a randomized trial comparing the treatment efficacy of Nivolumab versus chemotherapy in first line therapy of advanced non-small cell lung cancer based on the programmed death-ligand 1 expression. However, there was no strong correlation between treatment response and PD-L1 expression. Therefore, researchers performed a subanalysis to assess if the TMB could determine Nivolumab treatment response in 312 patients with evaluable TMB data. The results demonstrated that patients with a high mutation burden had a better progression free survival (9.7 vs 5.8 months; HR, 0.62) and objective response rate (46.8% vs 28.3%) compared with the control arm. These findings imply that tumor mutation burden may be considered as a biomarker for immunotherapy26.

Regarding TMB data, the CheckMate227 study is an open-label, phase 3 trial, that examined progression-free survival with nivolumab plus ipilimumab versus chemotherapy among patients with stage IV or recurrent NSCLC that was not previously treated with chemotherapy with a high tumor mutational burden (≥10 mutations per megabase). Median PFS among patients with a high tumor mutational burden was significantly longer with nivolumab plus ipilimumab than with chemotherapy, 7.2 months (95% confidence interval [CI], 5.5 to 13.2) versus 5.5 months (95% CI, 4.4 to 5.8) (HR, 0.58; 97.5% CI, 0.41 to 0.81; P<0.001)<sup>27</sup>.



Further understanding the factors associated with increased TMB is important for better understanding this key driver of cancer progression and for understanding the molecular mechanisms which lead to TMB.

Unlike the majority of genetic panels used within the standard of practice in oncology, even those using Next Generation Sequencing (NGS), Foundation Medicine <sup>®</sup> (FMI) is a "Comprehensive Genomic Profiling" test, able to detect all cancer-relevant genes with all classes of alterations across the entire coding region, being also a validated performance<sup>36</sup>. Moreover, is a hybridization capture-based NGS method which, contrary to the more common Hot Spot Multi-gene panels, do not miss any relevant gene or genetic alteration<sup>37</sup>. Besides, FMI has two formats, both of them validated in top tier peer-reviewed journal: "FoundationOne <sup>®</sup>" for solid tumors<sup>37</sup>. Finally, current service has been implemented for detection of Microsatellite Instability (MSI) and Tumor Mutational Burden (TMB).

Based on the above synergistic effects, Atezolizumab plus Bevacizumab might provide significant TMB selected NSCLC patients. For this reason, the Fundación GECP finds of great interest the following protocol: A phase 2 study evaluating the efficacy of Atezolizumab in combination with Bevacizumab as first line therapy for advanced or metastatic high-intermediate TMB (TMB≥10 mutations/MB analyzed in tumor or TMB≥16 analyzed in blood) non-squamous NSCLC patients.

# **Objectives and endpoints:**

# **Primary objective:**

 To evaluate the efficacy of Atezolizumab in combination with Bevacizumab as measured by Progression Free Survival (PFS) at 12 months according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.

# Secondary objectives:

- To evaluate the ORR of Atezolizumab in combination with Bevacizumab as measured by investigator-assessed overall response rate (ORR) according to RECIST v1.1.
- To evaluate the efficacy of Atezolizumab in combination with Bevacizumab as measured by investigator-assessed duration of response (DOR) according to RECIST v1.1.
- To evaluate the efficacy of Atezolizumab in combination with Bevacizumab as measured by investigator-assessed time to response (TTR) according to RECIST v1.1.
- To evaluate the efficacy of Atezolizumab in combination with Bevacizumab as measured by investigator-assessed ORR, PFS and DOR according to immune-related response criteria; irRC.
- To evaluate the efficacy of Atezolizumab in combination with Bevacizumab as measured by investigator ORR, PFS and DOR according to immune-related response criteria (irRC) in patients with TMB ≥16 mutations/MB.
- To evaluate the PFS rate at 1 and 2 years of Atezolizumab in combination with Bevacizumab.
- To evaluate the OS rate at 1 and 2 years of Atezolizumab in combination with Bevacizumab.



- To evaluate ORR and PFS according PD-L1 expression of Atezolizumab in combination with Bevacizumab.
- To evaluate the safety and tolerability of Atezolizumab in combination with Bevacizumab.
- To evaluate patient-reported outcomes (PROs) of lung cancer symptoms, patient functioning, and health-related quality of life (HRQoL) as measured by the European Organisation for Research and treatment of Cancer (EORTC) Quality-of-life Questionnaire Core 30 (QLQ C30) and its Lung Cancer Module (QLQ LC13) of Atezolizumab in combination with Bevacizumab.

# **Exploratory Objectives**

# Foundation one:

- To determine the tumor mutational burden (TMB) and determine its association with all 4 types of genomic alteration (Indels, mutation, CNV, rearrangement) in 324 tumor related genes, MSI and determine by FoundationOne CDx™ (F1CDx), and other biomarkers such as tumor PD-L1 expression.
- To investigate genomics alteration change measure in blood after progression measured with FoundationOne®Liquid, in respect with genomics alteration measure by FoundationOne CDx™ (F1CDx) in tissue including genomics signatures (MSI and TMB) at progression.
- To evaluate the clinical utility of the TMB results/reports in patients with TMB<10, mutations/MB describing druggable alterations or driver mutation that influence treatment selection.
- To evaluate overall survival (OS) and ORR of atezolizumab in combination with bevacizumab based on the TMB analysis in blood and in tumor)

# Additional pharmacogenomic exploratory analysis:

- To evaluate the basal peripheral blood TCR and BCR repertoire and their changes during treatment, as well as, their correlation with clinical variables associated with treatment efficacy (ORR, PFS, OS, DOR).
- To study the levels of peripheral blood immune cells and soluble factors from plasma samples considering their changes during treatment, as well as, their correlation with clinical variables associated with treatment efficacy (ORR, PFS, OS, DOR).
- To determine the pre-treatment fecal microbiome of all patients included in the study and its predictive value in terms of ORR, PFS, OS and DOR.

# **Eligibility criteria:**

# Inclusion criteria:

- 1. Male or female, aged ≥ 18 years old
- 2. ECOG performance status of 0 or 1.



- 3. Histologically or cytologically confirmed, Stage IIIB IV non-squamous NSCLC according to 8<sup>th</sup> version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology
- 4. No prior treatment for Stage IIIB IV non-squamous NSCLC.
- 5. Patients who have received prior neo-adjuvant, adjuvant chemotherapy, radiotherapy, or chemo-radiotherapy with curative intent for non-metastatic disease must have experienced a treatment-free interval of at least 6 months from enrollment since the last chemotherapy, radiotherapy, or chemo-radiotherapy.
- 6. Patients with a treated asymptomatic CNS metastasis are eligible, provided they meet all of the following criteria:
  - a. Only supratentorial and cerebellar metastases allowed (i.e., no metastases to midbrain, pons, medulla or spinal cord).
  - b. No ongoing requirement for corticosteroids as therapy for CNS disease.
  - c. No stereotactic radiation within 7 days or whole-brain radiation within 14 days prior to enrollment.
  - d. No evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study.

Patients with new asymptomatic CNS metastases detected at the screening scan must receive radiation therapy and/or surgery for CNS metastases. Following treatment, these patients may then be eligible without the need for an additional brain scan prior to inclusion, if all other criteria are met.

- 7. Patients with high-intermediate Tumor Mutational Burden analyzed by Foundation Medicine (≥10 mutations/ MB) performed by a Foundation Medicine laboratory on previously obtained archival tumor tissue or tissue obtained from a biopsy at pre-screening (sample must fulfil minimal sample requirements of 20% tumor cellularity and a minimum surface of 25mm²). TMB≥16 mutations/ MB is required if the analysis is performed in blood sample.
- 8. Measurable disease, as defined by RECIST v1.1.
  - Previously irradiated lesions can only be considered as measurable disease if disease progression has been unequivocally documented at that site since radiation and the previously irradiated lesion is not the only site of disease.
- 9. Adequate hematologic and organ function defined by the following laboratory results obtained within 14 days prior to enrollment:
  - Neutrophils ≥ 1500 cells/µL without granulocyte colony-stimulating factor support.
  - Lymphocyte count ≥ 500/μL.
  - Platelet count ≥ 100,000/μL without transfusion.
  - Haemoglobin ≥ 9.0 g/dL. Patients may be transfused to meet this criterion.
  - INR or aPTT ≤ 1.5 × upper limit of normal (ULN). This applies only to patients who are
    not receiving therapeutic anticoagulation; patients receiving therapeutic
    anticoagulation should be on a stable dose.
  - AST, ALT, and alkaline phosphatase ≤ 2.5 × ULN, with the following exceptions:
     Patients with documented liver metastases: AST and/or ALT ≤ 5 × ULN.

     Patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 × ULN.
  - Serum bilirubin ≤ 1.25 × ULN. Patients with known Gilbert disease who have serum bilirubin level ≤ 3 × ULN may be enrolled.
  - Serum creatinine ≤ 1.5 × ULN or creatinine clearance of ≥45ml/min (based on the Cockcroft Gault formula).



- 10. All patients are notified of the investigational nature of this study and signed a written informed consent in accordance with institutional and national guidelines, including the Declaration of Helsinki prior to any trial-related intervention.
- 11. For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate (< 1% per year) when used consistently and correctly, and to continue its use for 5 months after the last dose of Atezolizumab and/or 6 months after the last dose of Bevacizumab, whichever is later. Such methods include: combined (oestrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide, intrauterine device (IUD): intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.
- 12. For male patients with female partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate [< 1% per year] when used consistently and correctly, and to continue its use for 6 months after the last dose of Bevacizumab. Male patients should not donate sperm during this study and for at least 6 months after the last dose of Bevacizumab.
- 13. Oral contraception should always be combined with an additional contraceptive method because of a potential interaction with the study drugs. The same rules are valid for male patients involved in this clinical study if they have a partner of childbirth potential. Male patients must always use a condom.
- 14. Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 8 days prior to initiation of study drug.

# **Exclusion criteria:**

Cancer-Specific Exclusions:

- 1. Patients with a sensitizing mutation or an amplification in the epidermal growth factor receptor (EGFR) gene.
- 2. Patients with an anaplastic lymphoma kinase (ALK) fusion oncogene.
- 3. Patients with an STK-11 Ligand alteration.
- 4. Patients with MDM2 amplification.
- 5. Patients with ROS1 translocations.
- 6. Active or untreated CNS metastases as determined by CT or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments.
- 7. Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to enrollment.
- 8. Leptomeningeal disease.
- 9. Uncontrolled tumor-related pain.

Patients requiring pain medication must be on a stable regimen at study entry. Symptomatic lesions amenable to palliative radiotherapy (e.g., bone metastases or metastases causing nerve impingement) should be treated prior to initiation of study drug.



Patients should be recovered from the effects of radiation. There is no required minimum recovery period.

Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for locoregional therapy, if appropriate, prior to initiation of study drug.

- 10. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).
  - Patients with indwelling catheters (e.g., PleurX®) are allowed.
- 11. Uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or Ca > 12 mg/dL or corrected serum calcium > ULN).
- 12. Malignancies other than NSCLC within 5 years prior to enrollment, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous-cell skin cancer, localized prostate cancer treated with radiotherapy or surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent).

# **General Medical Exclusions:**

- 13. Women who are pregnant, lactating, or intending to become pregnant during the study.
- 14. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
- 15. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the Atezolizumab formulation.
- 16. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study.

Patients with controlled Type 1 diabetes mellitus on a stable dose of insulin regimen are eligible for this study.

Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

- Rash must cover less than 10% of body surface area (BSA).
- Disease is well controlled at baseline and only requiring low-potency topical steroids.
- No acute exacerbations of underlying condition within the previous 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high-potency or oral steroids).
- 17. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.



History of radiation pneumonitis in the radiation field (fibrosis) is permitted.

- 18. Positive test for HIV. All patients will be tested for HIV prior to inclusion into the study; patients who test positive for HIV will be excluded from the clinical study.
- 19. Patients with active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C.

Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible only if they are negative for HBV DNA (vaccinated patients are excluded). Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA.

- 20. Active tuberculosis.
- 21. Severe infections within 4 weeks prior to be included in the study, including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
- 22. Received therapeutic oral or IV antibiotics within 2 weeks prior to be included in the study.

  Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible.
- 23. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction, or cerebrovascular accident within 3 months prior to inclusion, unstable arrhythmias, or unstable angina.

Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.

- 24. Major surgical procedure other than for diagnosis within 28 days prior to inclusion or anticipation of need for a major surgical procedure during the course of the study.
- 25. Prior allogeneic bone marrow transplantation or solid organ transplant.
- 26. Administration of a live, attenuated vaccine within 4 weeks before inclusion or anticipation that such a live attenuated vaccine will be required during the study.
- 27. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications.
- 28. Patients with illnesses or conditions that interfere with their capacity to understand follow and/or comply with study procedures.

# **Exclusion Criteria Related to Medications:**

- 29. Any approved anti-cancer therapy, including hormonal therapy, within 3 weeks prior to initiation of study treatment.
- 30. Treatment with any other investigational agent with therapeutic intent within 28 days prior to initiation of study treatment.
- 31. Treatment with systemic immunosuppressive medications (including but not limited to corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to inclusion.

Patients who have received acute, low-dose (≤ 10 mg oral prednisone or equivalent), systemic immunosuppressant medications may be enrolled in the study.



The use of corticosteroids ( $\leq$  10 mg oral prednisone or equivalent) for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency is allowed.

# Exclusions Related to Bevacizumab:

32. Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg).

Anti-hypertensive therapy to achieve these parameters is allowable.

- 33. Prior history of hypertensive crisis or hypertensive encephalopathy.
- 34. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to inclusion.
- 35. History of haemoptysis (≥ one-half teaspoon of bright red blood per episode) within 1 month prior to inclusion.
- 36. Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation).
- 37. Current or recent (within 10 days of inclusion) use of aspirin (> 325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol.
- 38. Current use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes that has not been stable for > 2 weeks prior to inclusion.

The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks prior to inclusion.

Prophylactic anticoagulation for the patency of venous access devices is allowed, provided the activity of the agent results in an INR  $< 1.5 \times ULN$  and aPTT is within normal limits within 14 days prior to inclusion.

Prophylactic use of low-molecular-weight heparin (i.e., enoxaparin 40 mg/day) is permitted.

- 39. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to the first dose of Bevacizumab.
- 40. History of abdominal or tracheoesophageal fistula or gastrointestinal perforation within 6 months prior to inclusion.
- 41. Clinical signs of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding.
- 42. Evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
- 43. Serious, non-healing wound, active ulcer, or untreated bone fracture.
- 44. Proteinuria, as demonstrated by urine dipstick or > 1.0 g of protein in a 24-hour urine collection.

All patients with  $\geq$  2+ protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection and must demonstrate  $\leq$  1 g of protein in 24 hours.

- 45. Known sensitivity to any component of Bevacizumab.
- 46. Clear tumor infiltration into the thoracic great vessels is seen on imaging.
- 47. Clear cavitation of pulmonary lesions is seen on imaging.



# **Treatment:**

Atezolizumab: 1200mg, IV infusion Bevacizumab: 15 mg/kg, IV infusion

The treatment will start within 1-5 days from enrollment. The treatment will be administered at 21-day intervals (3 weeks ±3days). On Day 1 of each cycle, all eligible patients will receive drug infusions in the following order:

Atezolizumab → Bevacizumab

Atezolizumab may continue beyond disease progression per RECIST v1.1 until loss of clinical benefit, unacceptable toxicity, patient or physician decision to discontinue, or death. If the principal investigator would like to continue beyond progression a permission from the trial chair/sponsor have to be granted. For all patients, tumor response data collection will continue until disease progression, even if the patient stops study treatment prior to disease progression.

Bevacizumab will be administered until progression disease, unacceptable toxicity, patient or physician decision to discontinue or death.

# Statistical considerations:

The primary endpoint is Progression Free Survival (PFS) at 12 months according to Response Evaluation Criteria in Solid tumors (RECIST) v1.1.

For one arm, we estimate to achieve a PFS at 12 months of 40% (vs 18% from Chemotherapy, previous published studies), with a 90% power and alpha 5%, one-sided test. The test statistic for survival probability is based on the non-parametric estimate of the survival distribution. Additionally, estimating a 10% of errors, withdrawals or others, it will be necessary to recruit 40 patients in order to get the study objectives

If the withdrawals are higher than 5%, so that in order to reach the proposed sample size, if a patient initially enrolled in the study does not fulfil the inclusion criteria, they will be replaced by a new one subject that fulfil them, this replacement will ensure that the sample size will be the one calculated initially.

# Data analysis and statistical methods

A descriptive analysis will be made of the variables calculating absolute and relative frequencies of qualitative variables and mean (standard deviation) or median (25 and 75 percentiles), minimum and maximum values for quantitative variables.

For the primary endpoint analysis, survivor function estimated by Kaplan-Meier method will be used, as well as the survival curves. The 95% confidence interval will be estimated.



**Translational research:** 

For the bivariate analysis, appropriate parametric and nonparametric tests will be used depending on whether the data are normally or non-normally distributed. For comparison of quantitative variables, Student's t test for independent data, the Mann-Whitney U test, analysis of variance or the Kruskal-Wallis H test will be used.

**Total trial duration:** 4.5 years (1.5 years of recruitment, approximately 1.5 years of treatment and 1.5 years of follow up)



# 2. Trial schedule

| Pre-Screening | Screening/<br>Baseline<br>(-28 days before<br>enrollment) | Bevacizumab and<br>Atezolizumab<br>Cycles <sup>16</sup> | Atezolizumab Cycles (beyond progression disease) <sup>17</sup> | End of<br>Treatment <sup>18</sup> | Follow up <sup>19</sup> |
|---|---|---|---|---|---|
| | ı | | | | |
| | ı | | | | |
| | ı | | | | |
| | 1 | | | | |
| | - | | | | |



| T |
|---|



| 8 |
|---|



# 3. Background and rationale

# 3.1. Disease background and treatments in advanced NSCLC patients

Lung cancer is the leading cause of cancer-related death in industrialized countries<sup>1</sup>. Non-small cell lung cancer (NSCLC) accounts for 85% of cases of lung cancer and is categorized into a variety of histological subtypes being non-squamous tumors the most common subtype<sup>2</sup>.

Despite recent improvements in treatment, the prognosis for patients with advanced NSCLC remains dismal, with a median OS of approximately 12.5 months<sup>3</sup>.

Inhibition of programmed cell death protein-ligand 1/programmed cell death protein 1 (PD-L1/PD-1) signalling has been shown to induce durable responses in some patients with different tumors, and expression of PD-L1 by tumor cells (TCs) in several tumor types (including NSCLC) correlates with response to therapy<sup>4</sup>. Immunotherapy has demonstrated that therapies focused on enhancing T-cell responses against cancer may result in a significant survival benefit in patients with Stage IV cancer<sup>5,6,7</sup>.

Immunotherapeutic targeting of PD-L1 or PD-1 is revolutionizing the treatment of metastatic NSCLC. Currently, two anti-PD-1 therapeutic antibodies (Pembrolizumab and Nivolumab) and one anti-PD-L1 (Atezolizumab) have been approved for NSCLC treatment. Both agents are recommended as second-line agents in advanced NSCLC after prior progression on platinum-containing chemotherapy.

Atezolizumab is a humanized anti-PD-L1 monoclonal antibody that inhibits its interaction with its receptors, PD-1 and B7.1 (CD80, B7-1), reinvigorating anticancer immunity. The OAK study evaluated the efficacy of Atezolizumab compared to Docetaxel in 1.225 patients previously treated with locally-advanced or metastatic NSCLC. The PD-L1 targeted therapy by Atezolizumab resulted in a clinically relevant improvement of overall survival *versus* Docetaxel regardless of PD-L1 expression or histology, with a favourable safety profile. The median OS in this study was 13.8 months (95% CI 11.8-15.7) in the Atezolizumab arm compared to 9.6 months (95% CI 8.6-11.2) in the Docetaxel arm (HR=0.73, 95% CI 0.62-0.87; p=0.0003)<sup>8</sup>.

The GO28625 (NCT01846416, FIR) phase 2 study enrolled 137 PD-L1-selected NSCLC patients regardless previous treatments. The primary analysis for efficacy-evaluable patients, confirmed ORR after the first-line treatment with Atezolizumab was 28.6% (95% CI: 3.7-71.0) in IHC TC3 or IC3 patients and 25.8% (95% CI: 11.9-44.6) in IHC TC2/3 or IC2/3 patients<sup>9</sup>.

The efficacy and safety of Atezolizumab was also evaluated in another phase 2 single-arm study where 142 PD-L1-selected advanced NSCLC patients (NCT02031458, BIRCH) were treated with Atezolizumab monotherapy. The primary endpoint ORR in the ITT population was 25%, in TC3 or IC3 subgroup was 34% and 18% in TC2 and IC2. Median PFS and OS for the entire population were 7.3 and 23.5 months respectively. These results indicate that Atezolizumab monotherapy has durable efficacy in the first line setting <sup>10</sup>.



Currently, first-line treatment for advanced NSCLC without presence of genetic aberrations, such as sensitizing mutations of epidermal growth factor receptor (EGFR) or translocations of anaplastic lymphoma kinase (ALK), are chemotherapy and Pembrolizumab, approved based on KEYNOTE-024 study. This study randomized patients with advanced NSCLC and PD-L1 expression (at least 50% of tumor cells), showing median progression-free survival (PFS) of 10.3 months (95% CI 6.7-not reached) versus 6.0 months (95% CI 4.2-6.2) (HR 0.50; 95% CI 0.37-0.68; P<0.001) for the Pembrolizumab and chemotherapy groups respectively<sup>11</sup>.

Currently there is a clinical trial (NCT02409342, IMpower110) of Atezolizumab as first line monotherapy in PD-L1 selected NSCLC patients that is expected to add the first line approval to Roche's portfolio. Thus, all the above data support the rational of cancer immunotherapy in first line PD-L1 positive NSCLC<sup>12</sup>. In addition, there is a growing body of evidence that suggests that proangiogenic factors can modulate the immune response and may serve as mechanisms of scape. Therefore, the combination of cancer immunotherapy with antiangiogenic agents makes sense.

The vascular endothelial growth factor (VEGF) is the most important pro-angiogenic protein and a key regulator of physiological angiogenesis. It is also implicated in pathological angiogenesis associated with tumor growth. Indeed, increased levels of VEGF have been found in lung cancer; moreover, the overexpression of VEGF is associated with a poor prognosis<sup>13,14</sup>. Actually, VEGF plays a role in cancer immune evasion through modification of the endothelial cells in the tumor microenvironment, where VEGF may reduce lymphocyte adhesion and migration from vessels to the tumor site contributing to decreased immune cell recruitment<sup>15</sup>. Given the immunosuppressive role of VEGF and angiogenesis within tumors, it is not surprising that there is evidence supporting how antiangiogenic agents stimulate the immune response and enhance the efficacy of immunotherapies<sup>16</sup>.

Recent findings indicating an intertwined regulation of VEGF signalling and immunosuppression in the tumor microenvironment suggest that the combination of anti-VEGF agents and immune checkpoint blockade could have synergistic antitumor activity, along with favourable tolerability<sup>16</sup>.

Bevacizumab is a recombinant, humanized therapeutic anti-VEGF antibody that inhibits tumor angiogenesis which may correct the immunosuppressive function exerted by VEGF, increasing the infiltration of T effector cells in cancer<sup>17</sup>.

So far, the more advanced studies to address the combination of cancer immunotherapy (CIT)-antiangiogenic agents such as Bevacizumab, there is a phase 3 study of Paclitaxel, Carboplatin, Bevacizumab and Atezolizumab (NCT02366143, IMpower150). IMpower150 is the first phase III immunotherapy-based combination study to demonstrate a statistically significant and clinically meaningful improvement in PFS in all-comer 1L NSQ mNSCLC, providing a potential new standard of care for patients, showing a median PFS of 8.3 moths vs 6.8 moths (HR 0.62; 95% CI: 0.52, 0.74; P < 0.0001) for the Atezolizumab, chemotherapy and Bevacizumab arm (ABCP) and Carboplatin, Paclitaxel and Bevacizumab arm (BCP) respectively. In terms of PFS 12 months the results were 37% in the Atezolizumab arm vs 18% un the CT + Bevacizumab arm. Median overall survival among the patients was longer in the ABCP group than in the BCP group (19.2 months vs. 14.7 months; hazard ratio for death, 0.78; 95% CI, 0.64 to 0.96; P = 0.02)<sup>18</sup>.



The phase 3 study of Atezolizumab in combination with Bevacizumab compared to Sunitinib single agent (IMmotion151), as first-line therapy in untreated metastatic Renal Cell Carcinoma (RCC) patients. This clinical trial showed a significant benefit of 3.5 months in the PFS favouring the CIT-Bevacizumab combination (11.2 m vs. 7.7 m) with a tolerable safety profile in PD-L1+ patients<sup>19</sup>.

These data confirm the role of Bevacizumab as an immune modulating agent that may provide a successful combination strategy in different tumor types.

Increased mutation rate is a well-characterized feature of human cancer. Abnormal activity in several cellular pathways, including DNA damage repair and DNA replication, can increase the overall rate of somatic mutations in tumors, as can exposure to mutagens such as ultraviolet light and tobacco smoke<sup>20</sup>. Defects in DNA damage repair lead to the accumulation of mutations caused by replicative errors and environmental damage<sup>21</sup>.

The core DNA mismatch repair protein complex is composed of two cooperative dimers: the PMS2 protein dimerizes with MLH1 to form the complex MutL-alpha, which cooperates with the MSH2-MSH6 dimer, MutS-alpha, to repair single base pair mismatches and small insertion—deletion loops<sup>22</sup>. PMS2 promoter mutations are present in ~10% of melanoma samples and ~8% of squamous cell carcinomas<sup>23</sup>.

Perturbations in mismatch repair gene expression, both loss and overexpression, can be deleterious to genomic stability, and loss of function mutations in mismatch repair pathway genes are known to correlate with high Tumor Mutational Burden (TMB) in tumors, overall mutations in these genes accounted for less than 10% of cases with high TMB<sup>23</sup>.

As such, tumors with defective DNA repair mechanisms are more likely to benefit from immunotherapy. DNA replication is another key pathway in which defects can lead to increased somatic mutation rate.

Loss of function mutations in TP53 are very common in cancer and are a somatic marker of elevated mutation rate<sup>24</sup>. Mutations in a number of other genes have also been linked to increase TMB. KRASmutant lung cancers account for approximately 25% of non-small cell lung carcinomas, thus representing an enormous burden of cancer worldwide. KRAS mutations are clear drivers of tumor growth and are characterized by a complex biology involving the interaction between mutant KRAS, various growth factor pathways, and tumor suppressor genes. KRAS mutations are classically associated with a significant smoking history<sup>25</sup>. Then, it is an emerging biomarker for response to immunotherapy. The CheckMate 026 trial is a randomized trial comparing the treatment efficacy of Nivolumab versus chemotherapy in first line therapy of advanced non-small cell lung cancer based on the programmed death-ligand 1 expression. However, there was no strong correlation between treatment response and PD-L1 expression. Therefore, researchers performed a sub analysis to assess if the TMB could determine Nivolumab treatment response in 312 patients with evaluable TMB data. The results demonstrated that patients with a high mutation burden had a better progression free survival (9.7 vs 5.8 months; HR, 0.62) and objective response rate (46.8% vs 28.3%) compared with the control arm. These findings imply that tumor mutation burden may be considered as a biomarker for immunotherapy<sup>26</sup>.

Regarding TMB data, the CheckMate227 study is an open-label, phase 3 trial, that examined



progression-free survival with nivolumab plus ipilimumab versus chemotherapy among patients with stage IV or recurrent NSCLC that was not previously treated with chemotherapy with a high tumor mutational burden (≥10 mutations per megabase). Median PFS among patients with a high tumor mutational burden was significantly longer with nivolumab plus ipilimumab than with chemotherapy, 7.2 months (95% confidence interval [CI], 5.5 to 13.2) versus 5.5 months (95% CI, 4.4 to 5.8) (HR, 0.58; 97.5% CI, 0.41 to 0.81; P<0.001)<sup>27</sup>.

Unlike the majority of genetic panels used within the standard of practice in oncology, even those using Next Generation Sequencing (NGS), Foundation Medicine <sup>®</sup> (FMI) is a "Comprehensive Genomic Profiling" test, able to detect all cancer-relevant genes with all classes of alterations across the entire coding region, being also a validated performance<sup>36</sup>. Moreover, is a hybridization capture-based NGS method which, contrary to the more common Hot Spot Multi-gene panels, do not miss any relevant gene or genetic alteration<sup>37</sup>. Besides, FMI has two formats, both of them validated in top tier peer-reviewed journal: "FoundationOne <sup>®</sup>" for solid tumors<sup>37</sup>. Finally, current service has been implemented for detection of Microsatellite Instability (MSI) and Tumor Mutational Burden (TMB).

# 3.2. Immunotherapy

Several studies in patients with NSCLC suggested an association of increased immune cell infiltration into tumors with improved survival. In recent years, improved identification of antigenic targets, the addition of immunoadjuvants, and the production of more efficient delivery systems have resulted in more efficient vaccines, able to elicit a potent immune response, leading to the development of immunotherapy for the treatment of NSCLC<sup>28</sup>.

# 3.3. Background on Atezolizumab

Atezolizumab (MPDL3280A) is a humanized immunoglobulin (Ig) G1 monoclonal antibody consisting of two heavy chains (448 amino acids) and two light chains (214 amino acids) and is produced in Chinese hamster ovary cells. Atezolizumab was engineered to eliminate Fc-effector function via a single amino acid substitution on position 298 of the heavy chain, which results in a non-glycosylated antibody that has minimal binding to Fc receptors and prevents Fc-effector function at expected concentrations in humans.

Atezolizumab blocks the interaction between Programmed death-ligand 1 (PD-L1 or B7-H1) and Programmed death-1 (PD-1) and B7.1 (CD80), both of which are negative regulators of T-lymphocyte activation<sup>29</sup>. Binding of PD-L1 to its receptors suppresses T-cell migration, proliferation and secretion of cytotoxic mediators and restricts tumor cell killing. Blocking PD-L1 enhances anticancer immunity by restoring antitumor T-cell activity and T-cell priming.

# **Clinical Pharmacokinetics and Immunogenicity**

On the basis of available preliminary PL data (0.03-20 mg/kg), atezolizumab appeared to show linear pharmacokinetics at doses  $\geq$  1mg/kg. For the 1-mg/kg and 20-mg/kg dose groups, the mean apparent clearance and the mean volume of distribution under steady-state conditions had a range of 3.11 to 4.14 mL/kg and 48.1 to 67.0 mL/kg, respectively, which is consistent with the expected profile of an lgG1 antibody in humans.



The development of anti-therapeutic antibodies (ATAs) has been observed in patients in all dose cohorts and was associated with changes in pharmacokinetics for some patients in the lower dose cohorts (0.3, 1, and 3 mg/kg). The development of detectable ATAs has not had a significant impact on pharmacokinetics for doses from 10 to 20 mg/kg. Patients dosed at the 10-, 15- and 20-mg/kg dose levels have maintained the expected target trough levels of drug despite detection of ATAs. To date, no clear relationship among ATAs detection and adverse events or infusion reactions or efficacy has been observed.

# **Summary of Nonclinical Studies**

The nonclinical strategy of the atezolizumab program was to demonstrate in vitro and in vivo activity, to determine in vivo pharmacokinetic (PK) behaviour, to demonstrate an acceptable safety profile and to identify a Phase I starting dose. The safety, pharmacokinetics and toxicokinetics of atezolizumab were investigated in mice and cynomolgus monkeys to support intravenous (IV) administration and to aid in defining the appropriate starting dose in humans. The nonclinical pharmacokinetics and toxicokinetics observed for atezolizumab supported entry into clinical studies and were consistent with the anticipated pharmacologic activity of down-modulating the PD-L1/PD-1 pathway.

# **Summary of Clinical Studies**

Safety and efficacy data are summarized below from the following studies:

- Study PCD4989g: A Phase Ia, multicentre, first-in-human, open-label, dose-escalation study
  evaluating the safety, tolerability, immunogenicity, PK, exploratory pharmacodynamics and
  preliminary evidence of biologic activity of atezolizumab administered as a single agent by
  IV infusion every 3 weeks (q3w) to patients with locally advanced or metastatic solid
  malignancies or hematologic malignancies.
- Study GO28753 (POPLAR): A randomized, Phase II, open-label study assessing the clinical benefit of atezolizumab as a single agent versus docetaxel in PD-L1 unselected patients with locally advanced or metastatic NSCLC that has progressed during or following treatment with a platinum-containing regimen.
- Study OAK: A randomized, Phase III, open-label study assessing the clinical benefit of atezolizumab as a single agent versus docetaxel in PD-L1 unselected patients with previously treated advanced NSCLC that has progressed during or following treatment with a platinumcontaining regimen.
- Study GP28328: A Phase Ib study of the safety and pharmacology of atezolizumab administered with bevacizumab and/or with chemotherapy in patients with advanced solid tumors.

Currently atezolizumab is approved by FDA and EMA in patients with advanced NSCLC who progressed to previous therapies including platinum-based chemotherapy.



# Atezolizumab Single-Agent Safety Data on Patients with Advanced NSCLC

In the Phase I PCD4989g, in which atezolizumab was used as a single agent in patients with locally advanced or metastatic solid tumors or hematologic malignancies no maximum tolerated (MTD), no dose-limiting toxicities (DLTs) and no clear dose-related trends in the incidence of adverse events was determined. In this study, 520 out of 558 (93%) safety-evaluable patients experienced at least one adverse event, including 376 (67%) patients who experienced one treatment-related adverse event. Commonly reported events (≥10% of all patients) included fatigue, decreased appetite, nausea, pyrexia, constipation and cough. Grade 3-4 adverse events based on the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 [NCI CTCAE v4.0] were reported in 239 (43%) patients, of which 66 (12%) were considered related. Grade 3 and 4 adverse events considered related by the investigator included dyspnoea, pneumonitis, increased ALT, increase AST, increased GGT, lymphocyte count decreased, cardiac tamponade, asthenia, autoimmune hepatitis, pneumonia, influenza and hypoxia.

In the randomized Phase II POPLAR Study (GO28753), the frequency of patients who reported any adverse events regardless of attribution was 96% for both  $arms^{30}$ . A higher number of  $Grade \ge 3$  adverse events were observed in the docetaxel arm (53% vs 40%), explained mainly by the difference in adverse events due to bone marrow suppression. This difference was more evident in Grade 3-4 treatment-related adverse events (39% vs 11%). The most common atezolizumab Grade 3 adverse events were pneumonia (2%) and increased AST (2%). No atezolizumab-related Grade 4 adverse events were reported. Immune-related adverse events of any grade with atezolizumab were increased AST (4%), increased ALT (4%), pneumonitis (3%), colitis (1%) and hepatitis (1%). Fewer patients discontinued treatment with atezolizumab than with docetaxel (8% vs 22% respectively). There were six (4%) Grade 5 adverse events in atezolizumab were cardiac failure, pneumonia, ulcer haemorrhage, pneumothorax, pulmonary embolism and embolism.

In the randomized Phase III OAK Study, the frequency of patients who reported any adverse event regardless of attribution was similar in both arms: 94% in atezolizumab arm and 96% in docetaxel arm $^{31}$ . A higher number of Grade  $\geq 3$  adverse events were observed in the docetaxel arm (54%) compared with atezolizumab arm (37%). This difference was greater in Grade 3-4 treatment-related adverse events (43% vs 15%). The most common atezolizumab-related adverse events were fatigue (14%), nausea (9%), decreased appetite (9%) and asthenia (8%). Immune-related adverse events reported with atezolizumab included pneumonitis (1%), hepatitis (<1%) and colitis (<1%).

A pooled safety analysis conducted in 843 patients who received atezolizumab in 4 studies (PCD4989g [N = 76]; BIRCH [N = 520]; FIR [N = 105]; POPLAR [N = 142]) (Lukas et al. WCLC 2016). Twenty-seven (3%) of 843 patients had asymptomatic untreated brain metastases or stable previously treated brain metastases at baseline. The incidence of treatment-related neurological AEs was 4 (15%) in patients with baseline brain metastases, including the most common treatment-related AE of headache in 2 (7%) and 27 (3%) patients, respectively. The most common all-cause AEs



in patients with baseline brain metastases were fatigue, nausea, and vomiting (7 [26%] each). No treatment discontinuations occurred due to AEs.

# Atezolizumab in Combination with Platinum-Based Chemotherapy Safety Data on patients with Advanced NSCLC

The Study GP28328 is a Phase Ib study of atezolizumab in combination with bevacizumab or cytotoxic chemotherapy in patients with multiple tumor types including NSCLC, triple-negative breast cancer and colorectal cancer. Patients with advanced NSCLC were included in the following arms: Arm C (atezolizumab + carboplatin + paclitaxel), Arm E (atezolizumab + carboplatin + pemetrexed) and Arm E (atezolizumab + carboplatin + nab-paclitaxel). These combinations have been generally well tolerated and no DLTs have been reported during the dose-escalation stage in any study arm. A total of 141 of 144 (98%) patients reported at least one adverse event while receiving study drug. Most of these events were Grade 2 and 3 in severity. The five most commonly adverse events across the study arms (≥10%) included fatigue, nausea, diarrhoea, decreased appetite and pyrexia. The adverse events were consistent with the known safety profile of each agent and no additive effects were observed when atezolizumab was administered with chemotherapy.

# Atezolizumab Single-Agent Efficacy Data on Patients with Advanced NSCLC

In the Phase I PCD4989g Study, the efficacy evaluable population included 88 patients with locally advanced or metastatic NSCLC and represented a heavily pre-treated patient population (97% of the patients had received  $\geq$  2 prior systemic therapies and 77% had received  $\geq$  4 prior systemic therapies). Overall, responses were observed in 20 out of 88 (23%) patients with NSCLC and included responses in patients with squamous and non-squamous NSCLC (4 in 21 and 16 in 67 patients respectively).

In the POPLAR Study, the primary OS analysis was conducted when 173 deaths had occurred. Most patients had received one prior therapy (65%), had non-squamous histology (66%) and ECOG performance status of 1 (68%). Atezolizumab showed significant improvement in OS compared with docetaxel (12.6 vs 9.7 months; HR = 0.73, 95% CI 0.53-0.99; p = 0.04). OS benefit was associated with tumor PD-L1 overexpression. PFS was similar among both arms (2.7 vs 3 months respectively) and objective responses with atezolizumab were durable, with a median duration of 14.3 months compared with 7.2 months for docetaxel.

In the OAK Study, the primary efficacy analysis population comprised the first 850 patients. Most patients had received one prior therapy (75%), had non-squamous histology (74%) and ECOG performance status of 1 (63%). Atezolizumab showed significant improvement in OS compared with docetaxel (13.8 vs 9.6 months; HR = 0.73, 95% CI 0.62-0.87; p = 0.003). Based on the last data cut off with a minimum follow-up of 26 months, the 2-year OS rate in patients who received atezolizumab was 31% versus 21% in patients treated with docetaxel (Satouchi et al. WCLC 2017). Although the benefit in terms of OS was associated with tumor PD-L1 overexpression, patients with low or undetectable PD-L1 expression (ICO/TCO) also had improved OS with atezolizumab. A post-hoc



subgroup analysis showed that patients with stable previously treated BM also had significant benefit in OS and PFS from atezolizumab (Gadgeel et al. WCLC 2016).

# Atezolizumab in Combination with Platinum-Based Chemotherapy Efficacy Data on patients with Advanced NSCLC

In the Study GP28328, patients with advanced NSCLC received atezolizumab q3w in combination with platinum-based chemotherapy: carboplatin + paclitaxel (Arm C), carboplatin + pemetrexed (Arm D) and carboplatin + nab-paclitaxel (Arm E). All patients had histologically or cytologically documented Stage IIIB or IV or recurrent NSCLC and had not received prior chemotherapy for advanced disease. The median age was 65 years and 79% had non-squamous histology. In the first data cut off (February 10th 2015), 41 patients were evaluable for efficacy and the ORR in all three arms was 63%. In the last update of the study, 76 patients were evaluable for efficacy and the ORR according to the three arms was: Arm C (n=25) 46%; Arm D (n=25) 68%; Arm E (n=26) 36% (Liu et al. ASCO 2017). For patients treated with carboplatin + pemetrexed (Arm D), median PFS was 8.4 months (4.7-11) and OS rate at 12 months was 68%.

Refer to the local prescribing information for additional details on nonclinical and clinical studies.

# Rationale for Atezolizumab dose

The fixed dose of 1200 mg (equivalent to an average body weight-base dose of 15mg/kg) intravenously was selected on the basis of both nonclinical studies and available clinical data from Study PCD4989g. The target exposure for atezolizumab was projected on the basis of nonclinical tissue distribution data in tumor-bearing mice, target-receptor occupancy in the tumor, the observed atezolizumab interim pharmacokinetics and other factors.

Antitumor activity has been observed across doses from 1 mg/kg to 20 mg/kg. The MTD of atezolizumab was not reached and DLTs have been observed at any dose in Study PCD4989g. Currently available PK and ATA data suggest that the 15-mg/kg atezolizumab q3w regimen (or fixed-dose equivalent) for Phase II and Phase III studies would be sufficient to both maintain Ctrough  $\geq 6$  µg/mL and further safeguard against both interpatient variability and the potential effect of ATAs that may lead to subtherapeutic levels of atezolizumab relative to the 10-mg/kg atezolizumab q3w regimen.

In this trial, atezolizumab will be given as an intravenous fixed dose of 1200 mg every 3 weeks (q3w) until unacceptable toxicity or disease progression, as assessed by the investigator. Atezolizumab treatment could continue beyond disease progression if the investigator deems the patient to have clinical benefit.

# 3.4. Background on Bevacizumab

Bevacizumab is a recombinant humanized monoclonal IgG1 antibody that blinds to and inhibits the interaction of VEGF-A to its receptors (Flt-1 and KDR) on the surface of endothelial cells. The



interaction of VEGF with its receptors leads to endothelial cell proliferation and new blood vessel formation in *in vitro* models of angiogenesis.

Neutralising the biological activity of VEGF regresses the vascularisation of tumors, normalises remaining tumor vasculature, and inhibits the formation of new tumor vasculature, thereby inhibiting tumor growth.

Administration of Bevacizumab to xenotransplant models of colon in nude mice caused reduction of microvascular growth and inhibition of metastatic disease progression<sup>32,33</sup>.

Bevacizumab is indicated for the first line treatment of unresectable, locally advanced, recurrent or metastatic non-squamous non-small cell lung cancer. The recommended dose of bevacizumab is 15mg/Kg by IV infusion once every 3 weeks (21 days).

# 3.5. Rationale for trial design





3.6. Rationale for additional pharmacogenomic exploratory research (stool and blood samples)





# 4. Objectives and endpoints

# 4.1. Primary objective and endpoint

• To evaluate the efficacy of Atezolizumab in combination with Bevacizumab as measured by Progression Free Survival (PFS) at 12 months according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.

PFS after enrollment is defined as the time from enrollment to the first occurrence of disease progression or death from any cause, whichever occurs first.



# 4.2. Secondary objectives and endpoint

- To evaluate the Overall response rate (ORR) of Atezolizumab in combination with Bevacizumab as measured by investigator-assessed overall response rate (ORR) according to RECIST v1.1.
  - ORR defined as percentage of patients reaching complete or partial response.
- To evaluate the efficacy of Atezolizumab in combination with Bevacizumab as measured by investigator-assessed duration of response (DOR) according to RECIST v1.1.
  - DOR defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first.
- To evaluate the efficacy of Atezolizumab in combination with Bevacizumab as measured by investigator-assessed time to response (TTR) according to RECIST v1.1.
  - TTR defined as the time from the start of the treatment to the first objective tumor response observed for patients who achieved CR or PR.
- To evaluate the efficacy of Atezolizumab in combination with Bevacizumab as measured by investigator-assessed ORR, PFS and DOR according to immune-related response criteria; irRC.
- To evaluate the efficacy of Atezolizumab in combination with Bevacizumab as measured by investigator ORR, PFS and DOR according to immune-related response criteria (irRC) in patients with TMB ≥16.
- To evaluate the PFS rate at 1 and 2 years of Atezolizumab in combination with Bevacizumab.
- To evaluate the Overall Survival (OS) rate at 1 and 2 years of Atezolizumab in combination with Bevacizumab.
  - OS defined as the length of time from either the date of diagnosis or the start of the treatment that patients diagnosed with the disease are still alive.
- To evaluate ORR and PFS according PD-L1 expression of Atezolizumab in combination with Bevacizumab.
- To evaluate the safety and tolerability of Atezolizumab in combination with Bevacizumab.
   Occurrence and severity of adverse events, with severity determined by NCI CTCAE v5.0 criteria.
- To evaluate patient-reported outcomes (PROs) of lung cancer symptoms, patient functioning, and health-related quality of life (HRQoL) as measured by the European Organisation for Research and treatment of Cancer (EORTC) Quality-of-life Questionnaire



Core 30 (QLQ C30) and its Lung Cancer Module (QLQ LC13) of Atezolizumab in combination with Bevacizumab.

Change from baseline in quality of life, as assessed through use of the EORTC C30 and LC13 at baseline, at cycle 3, every 3 cycles until progression and at progression.

# 4.3. Exploratory objectives

# Foundation one:

- To determine the tumor mutational burden (TMB) and determine its association with all 4 types of genomic alteration (Indels, mutation, CNV, rearrangement) in 324 tumor related genes, MSI and determine by FoundationOne CDx™ (F1CDx), and other biomarkers such as tumor PD-L1 expression.
- To investigate genomics alteration change measure in blood after progression measured with FoundationOne®Liquid, in respect with genomics alteration measure by FoundationOne CDx™ (F1CDx) in tissue including genomics signatures (MSI and TMB) at progression.
- To evaluate the clinical utility of the TMB results/reports in patients with TMB<10, mutations/MB describing druggable alterations or driver mutation that influence treatment selection.
- To evaluate overall survival (OS) and ORR of atezolizumab in combination with bevacizumab based on the TMB analysis in blood and in tumor)

# Additional pharmacogenomic exploratory analysis:

- To evaluate the basal peripheral blood TCR and BCR repertoire and their changes during treatment, as well as, their correlation with clinical variables associated with treatment efficacy (ORR, PFS, OS, DOR).
- To study the levels of peripheral blood immune cells and soluble factors from plasma samples considering their changes during treatment, as well as, their correlation with clinical variables associated with treatment efficacy (ORR, PFS, OS, DOR).
- To determine the pre-treatment fecal microbiome of all patients included in the study and its predictive value in terms of ORR, PFS, OS and DOR.








 $<sup>^{</sup>st}$  If the submitted tumor sample is insufficient or not valid to evaluate the TMB, a blood sample can be sent instead .





| | _ |
|---|---|
| _ | |
| | = |
| | = |
| | = |
| | = |
| | = |
| | • |
| | • |
| | • |









| _ |
|---|
| - |









# 7. Patient pre-screening and enrollment

The patients will be eligible for the study after the tumor mutation burden (TMB) determination. This analysis will be done at the pre-screening phase of the study. The patient pre-screening form (appendix 8) has to be sent to the Fundación GECP headquarters scanned by email to the clinical monitor or by fax (+34 93 419 17 68). A pre-screening number will be assigned and returned to the participating hospital by fax or email. After the TMB determination if the patient has a TMB≥10 mut/MB analyzed in tumor or TMB≥16 analyzed in blood and fulfil all the eligibility criteria, the patient will be enrolled in the study.

Note that written informed consent has to be obtained from the patient prior to any trial-specific intervention. The patient has to sign a specific pre-screening informed consent to send the tumor block for pre-screening (TMB analysis). If the submitted tumor sample is insufficient or not valid and a biopsy is not feasible to be performed to evaluate the TMB, a blood sample can be sent instead.

A permission from the trial chair/sponsor must be requested in case no tumor sample is available for a possible patient and blood sample want to be sent to analyze the TMB.



If the patient has a TMB ≥10 analyzed in tumor TMB≥16 analyzed in blood then the patient will sign the Informed consent of the study.

This trial will use a web-based enrollment system (eCRF-Electronic Case Report Form). Each participating centre will access the system directly to enrol the patients.

Patient eligibility needs to be checked before enrollment of the patient in the Fundación GECP webbased system (eCRF). The dates of the patient signature of the Informed Consent of the study and the specific informed consent to pathology material submission for pre-screening are required to be filled in the eligibility checklist of the eCRF.

The treatment has to start preferably the date of enrollment or within 1-5 days from the date of enrollment.

# 8. Trial procedures

# 8.1. Overview of treatment sequence

#### 8.1.1. Pre-screening phase



#### 8.1.2. Screening/Baseline visit:



| _ |
|---|
| _ |
| _ |
| _ |
| • |
| _ |
| _ |
| _ |





# 8.1.3. Bevacizumab and Atezolizumab cycles



On Day 1 of each cycle, all eligible patients will receive drug infusions in the following order:

Atezolizumab: 1200mg, IV infusion
 Bevacizumab: 15 mg/kg, IV infusion

Patients should receive treatments according to the local standard of care and manufacturer's instruction. A suggested infusion times for treatment administration:

| | Atezolizumab | Bevacizumab |
|---------------|-------------------|------------------------|
| Infusion rate | Over 60 (±15) min | Over 90 (±15) min (for |
| in asion rate | (for the first | the first infusion); |



| infusion); | shortening to |
|------------------------|-------------------------|
| 30 (± 10) min for | 60 (± 10) then |
| subsequent | 30 (± 10) min for |
| infusions if tolerated | subsequent infusions if |
| illusions il tolerated | tolerated |

The following procedures must be performed on day 1 of each cycle (±3 days):

- 1. Physical examination, including: weight, ECOG, Temperature and blood pressure.
- 2. Blood pressure must be taken always before the drug administration. Blood pressure should be routinely measured before every infusion after a resting period of 10 min. If baseline record is performed more than 3 days before first study dose, they must be repeated on day 1 cycle 1.
- 3. Laboratory testing prior to each dose administration within 3 days prior to day 1 administration of each cycle. If baseline testing is performed more than 3 days before first study dose, they must be repeated on day 1 cycle 1:
  - **Hematology and coagulation**: WBC count, neutrophils, haemoglobin, platelet count, PT, INR and APTT.
  - Biochemistry: Ca, Mg, Na, K, Glucose, ALT, AST, LDH, total bilirubin, alkaline phosphatase, creatinine and clearance of creatinine calculated by Cockcroft-Gault formula, total protein, albumin, amylase, lipase.
  - Thyroid function: thyroid-stimulating hormone (TSH). Total or free T3 and total or free T4 must be analyzed if TSH result is out of ULN or LLN. It is required at cycle 2 and then every 2 cycles (more frequently if clinical indicated).
  - Pregnancy Tests: A serum or urine pregnancy testing is required at cycle 2 and then every 2 cycles (more frequently if required by local standard).
  - **Urine test**: A urine testing (dipstick is allowed) is required for proteinuria.
- 4. Adverse events: Changes from baseline symptoms (new or worsened clinically significant ones) should be recorded as adverse events on the Adverse Event form of the eCRF. For laboratory parameters, only grade 2 events will be reported as an AE. All the other events not related to laboratory values will be reported from grade 1.



- 5. Concomitant medications: Changes from baseline should be recorded on the eCRF.
- 6. Tumor assessment will be done every 12 weeks (± 7 days) from cycle 1 day 1. CT SCAN must be performed until progression disease or until last dose of Atezolizumab in case of continuing beyond progression. The CT SCAN schedule will be maintained even if a delay in administration occurs.
  - Chest and abdomen CT SCAN with oral/IV contrast (unless contraindicated) to determine measurable disease according to RECIST v1.1 (at least one lesion outside of irradiated areas that can be measured in at least one dimension as ≥ 10 mm, or ≥ 15 mm in case of lymph nodes).
  - A full-body PET-TAC, pelvis or the neck CT scan, MRI or CT brain and bone scans should be performed if clinically indicated.
- 7. PRO (QLQ30-LC13) must be performed always before dose administration, starting on day 1 of cycle 3 and then every 3 cycles. In the event of a delay in administration, the PROs schedule will be also delayed to be performed on day 1 of the specified cycles.
- 8. Pharmacogenomic exploratory analysis: blood samples will be drawn at:
  - First CT-scan evaluation (cycle 5 if there is no delay in treatment administration)
  - Second CT-scan evaluation (cycle 9 if there is no delay in treatment administration)
  - Fourth CT-scan evaluation (cycle 17 if there is no delay in treatment administration)
  - Sixth CT-scan evaluation (cycle 25 if there is no delay in treatment administration)
  - Progression disease, if it occurs during the bevacizumab + atezolizumab treatment

#### 8.1.4. Atezolizumab cycles (beyond progression):

Atezolizumab may continue beyond disease progression per RECIST v1.1 until loss of clinical benefit, unacceptable toxicity, patient or physician decision to discontinue, or death. If the principal investigator would like to continue beyond progression a permission from the trial chair/sponsor have to be granted.

Cycles will be administered every 3 weeks (±3 days). Patient will receive:

Atezolizumab: 1200mg, IV infusion



The following procedures must be performed on day 1 of each cycle (±3 days):

- 1. Physical examination, including: weight, ECOG, Temperature and blood pressure (always before the drug administration).
- 2. Laboratory testing prior to each dose administration within 72 hours prior to day 1 administration of each cycle:
  - Hematology and coagulation: WBC count, neutrophils, hemoglobin, platelet count, PT, INR and APTT.
  - Biochemistry: Ca, Mg, Na, K, Glucose, ALT, AST, LDH, total bilirubin, alkaline phosphatase, creatinine and clearance of creatinine calculated by Cockcroft-Gault formula, total protein, albumin, amylase, lipase.
  - Thyroid function: thyroid-stimulating hormone (TSH). Total or free T3 and total or free T4 must be analyzed if TSH result is out of ULN or LLN. It is required at cycle 2 and then every 2 cycles (more frequently if clinical indicated).
  - Pregnancy Tests: A serum or urine pregnancy testing is required at cycle 2 and then every 2 cycles (more frequently if required by local standard).
- 3. Adverse events: Changes from baseline symptoms (new or worsened clinically significant ones) should be recorded as adverse events on the Adverse Event form of the eCRF. For laboratory parameters, only grade 2 events will be reported as an AE. All the other events not related to laboratory values will be reported from grade 1.
- 4. Concomitant medications: Changes from baseline should be recorded on the eCRF.
- 5. Tumor assessment will be done every 12 weeks (± 7 days) from cycle 1 day 1. The CT SCAN schedule will be maintained even if a delay in administration occurs:
  - a. Chest and abdomen CT SCAN with oral/IV contrast (unless contraindicated) to determine measurable disease according to RECIST v1.1 (at least one lesion outside of irradiated areas that can be measured in at least one dimension as  $\geq$  10 mm, or  $\geq$  15 mm in case of lymph nodes).
  - b. A full-body PET-TAC, pelvis or the neck CT scan, MRI or CT brain and Bone scans should be performed if clinically indicated.

#### 8.1.5. End of treatment and first follow up visit



| _ |
|---------|
| <u></u> |





8.1.6. Follow up visits







#### 8.1.7. Quality of Life (QoL)

The quality of life (QoL) of patients will be assessed using EORTC QLQ-C30<sup>34</sup> and the lung cancer module (QLQ-LC13) questionnaires. The EORTC QLQ-C30<sup>34</sup> is a self-administered cancer specific questionnaire with multi-dimensional scales. It consists of both multi-item scales and single item measures, including five functioning domains, a global quality of life domain, three symptom domains and six single items. For each domain or single item measure a linear transformation will be applied to standardize the raw score to range between 0 and 100.

The QLQ-LC13 lung cancer module<sup>35</sup> includes questions assessing lung cancer-associated symptoms (cough, hemoptysis, dyspnea, and site-specific pain), treatment-related side effects (sore mouth, dysphagia, peripheral neuropathy and alopecia) and pain medication. The validity and reliability have been studied by the EORTC Study Group on Quality of Life. The EORTC QLQ-C30 and module will be scored according to the EORTC QLQ-C30 Scoring Manual and analyzed accordingly.

Changes of the quality of life scores while on treatment versus baseline will be examined using analysis and descriptive statistics. Specific time points will be checked to explore treatment side effect on patients QoL, and the longtime benefit of the study treatment.

Please see Sections 8.1.2, 8.1.3, 8.1.4, 8.1.5 and 8.1.6 to know the QoL tests schedules.

# 9. Investigational Medicinal Product

Atezolizumab and Bevacizumab are the Investigational Medicinal Products (IMP) used in this trial. Roche will provide the IMPs at no cost for this trial.

Complete details of the trial drug logistics, distribution, packaging, labelling, storage and handling as well as accountability are described in the *TELMA drug supply manual* that will be provided in the Pharmacy site file to all the participant sites.

**Description of the Investigational Medicinal Products** 



| 9.1. | Packaging and labelling |
|------|--------------------------------|
| 9.2. | Receipt and storage of the IMP |
| 9.3. | Unused trial drug supplies |



# 9.4. Treatment beyond trial closure

The Fundación GECP, the Sponsor of the TELMA trial, will offer continued access to the two Roche IMPs atezolizumab and bevacizumab free of charge to eligible participants in accordance with the Roche Global Policy on Continued Access to Investigational Medicinal Product.

# 9.4.1. Eligibility to receive atezolizumab and/or bevacizumab after study completion.

A participant will be eligible to receive Roche IMPs atezolizumab and/or bevacizumab after completing the study if all of the following conditions are met:

- The patient has received Roche IMPs atezolizumab and bevacizumab during study conduct, and
- The patient is still experiencing clinical benefit from Roche IMPs atezolizumab and/or bevacizumab at the time of study closure, and
- The patient has a life-threatening or severe medical condition and requires continued treatment with Roche IMPs atezolizumab and/or bevacizumab for their well-being, and
- There are no appropriate alternative treatments available to the participant, and
- The participant and their doctor comply with and satisfy any legal or regulatory requirements that apply to them.

#### 9.4.2. Safety reporting requirements beyond trial closure

The last dose of IMP administered before study closure shall be considered the last per protocol treatment administration. Any adverse events related to this last IMP dose and occurring within the time until the first off-study IMP administration (e.g. approximately 3 weeks) should be reported as described in Section 13. Adverse Events and Reporting. Beyond this timeline, any adverse events related to the IMP more than 30 days after the last administration of on-study IMP, should be reported by the treating physician to Roche and/or the appropriate body in accordance with local rules and regulations.

# 10. Trial treatments description

#### 10.1. ATEZOLIZUMAB





#### 11. Dose modifications criteria

Reasons for dose modifications, the supportive measures taken, and the outcomes will be documented in the patient's chart and recorded on the eCRF.

### 11.1. General Notes Regarding Dose Modification

- When several toxicities with different grades of severity occur at the same time, the dose modifications should be according to the highest grade observed.
- If, in the opinion of the investigator, a toxicity is considered to be due solely to one component of the study treatment (i.e., atezolizumab or bevacizumab) and the dose of that component is delayed or modified in accordance with the guidelines below, other components may be administered if there is no contraindication.
- When treatment is temporarily interrupted because of toxicity caused by bevacizumab or atezolizumab, the treatment cycles will be restarted such that the atezolizumab and bevacizumab infusions remain synchronized.

The investigator may use discretion in modifying or accelerating the dose modification guidelines described below depending on the severity of toxicity and an assessment of the risk versus benefit for the patient, with the goal of maximizing patient compliance and access to supportive care.

# 11.2. ATEZOLIZUMAB dose delay criteria



| 11.3. BEVACIZUMAB dose delay/reduction criteria |
|-------------------------------------------------|



| Management of bevacizumab related toxicities |
|----------------------------------------------|











| Surgery and wound healing complications |
|-----------------------------------------------------|
| Surgery and Wound nearing complications |
| 12. Prohibited and permitted concomitant treatments |



| Prohibited Concomitant Therapy |
|--------------------------------|
| Permitted Concomitant Therapy |



| _ | |
|---|------|
| - | |
| | - |
| | <br> |

# **Cautionary Concomitant Therapy**



# 13. Adverse events and reporting

#### 13.1. Definition of an Adverse Event (AE) and AE's reporting

| The main criterion for tolerability is the occurrence of toxicities and Adverse Events (AEs). |
|---|

An adverse event can therefore be any of the following:

Any unfavourable and unintended sign (including an abnormal laboratory finding) (see **NOTE 1** below), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Any new disease or exacerbation of an existing disease (a worsening in the character, frequency, or severity of a known condition), except events that are clearly consistent with the expected pattern of the disease progression. These data will be captured as efficacy assessment data only. If there is any uncertainty as to whether an event is due to disease progression, it should be reported as an adverse event.

Recurrence of an intermittent medical condition (e.g., headache) not present at baseline.

Any deterioration in a laboratory value or other clinical test (e.g., ECG, X-ray) that is associated with symptoms or leads to a change in study treatment or concomitant treatment or discontinuation from study drug.

Adverse events that are related to a protocol-mandated intervention, including those that occur prior to assignment of study treatment (e.g., screening invasive procedures such as biopsies).

Adverse events that occur during or within 24 hours after study drug administration and are judged to be related to study drug infusion should be captured as a diagnosis (e.g., "infusion-related reaction" or "anaphylactic reaction") on the Adverse Event eCRF. If a patient experiences both a local and systemic reaction to the same dose of study drug, each reaction should be recorded separately on the Adverse Event eCRF. Associated signs and symptoms should be recorded on the dedicated Infusion-Related Reaction eCRF.

A pre-existing medical condition should be recorded as an adverse event only if the frequency, severity, or character of the condition worsens during the study (e.g., "more frequent headaches").

**NOTE 1:** Abnormal laboratory and vital signs values:



A laboratory test result must be reported as an adverse event if it is a change from baseline and meets any of the following criteria:

Is accompanied by clinical symptoms,

Results in a change in study treatment (e.g., dosage modification, treatment interruption, or treatment discontinuation),

Results in a medical intervention (e.g., potassium supplementation for hypokalaemia) or a change in concomitant therapy,

Is clinically significant in the investigator's judgment.

If a clinically significant laboratory abnormality is not a sign of a disease or syndrome, the abnormality itself should be recorded on the Adverse Event eCRF, along with a descriptor indicating if the test result is above or below the normal range (e.g., "elevated potassium").

A vital sign result must be reported as an adverse event if it is a change from baseline and meets any of the following criteria:

Is accompanied by clinical symptoms,

Results in a change in study treatment (e.g., dosage modification, treatment interruption, or treatment discontinuation),

Results in a medical intervention or a change in concomitant therapy,

Is clinically significant in the investigator's judgment.

If a clinically significant vital sign abnormality is a sign of a disease or syndrome (e.g., high blood pressure), only the diagnosis (i.e., hypertension) should be recorded on the Adverse Event eCRF.

The finding of an elevated ALT or AST ( $> 3 \times$  baseline value) in combination with either an elevated total bilirubin ( $> 2 \times$  ULN) or clinical jaundice in the absence of cholestasis or other causes of hyperbilirubinemia is considered to be an indicator of severe liver injury. Therefore, investigators must report as an adverse event the occurrence of either of the following:

Treatment-emergent ALT or AST > 3  $\times$  baseline value in combination with total bilirubin > 2  $\times$  ULN (of which  $\geq$  35% is direct bilirubin),

Treatment-emergent ALT or AST > 3  $\times$  baseline value in combination with clinical jaundice.

This abnormal laboratory values related to the liver function should be recorded on the Adverse Event eCRF and reported immediately as a SAE (AESI).

The severity will be classified according to the NCI CTCAE Version 5.0. The CTCAE is available for downloading on the internet (see appendix 1).



The AE severity grade provides a qualitative assessment of the extent or intensity of an AE, as determined by the investigator or as reported by the patients. The severity grade does not reflect the clinical seriousness of the event, only the degree or extent of the affliction or occurrence (e.g., severe nausea, mild seizure), and does not reflect the relationship to study drug.

Severity grade for other adverse events not covered in the toxicity grading scale:

| 1 = Grade 1 | Mild |
|-------------|------------------|
| 2 = Grade 2 | Moderate |
| 3 = Grade 3 | Severe |
| 4 = Grade 4 | Life-threatening |
| 5 = Grade 5 | Fatal |

However, depending on the SAE term, there is some AE that do not have all the grades (e.g., the SAE term Alopecia only has the Grade 1 and 2).

The causal relationship to study drug is determined by the physician and should be used to assess all AE. The casual relationship can be one of the following:

**<u>Related</u>**: There is a reasonable causal relationship between study drug administration and the AE.

**Not related**: There is not a reasonable causal relationship between study drug administration and the AE.

The term "reasonable causal relationship" means there is evidence to suggest a causal relationship.

About the AEs that have to be recorded in the eCRF note that:

- Baseline symptoms will be recorded on the eCRF and changes and updates in grade as well as resolution of an AE during treatment have to be reported,
- An AE has to be reported for each SAE notified,
- AEs should not be reported in a narrative description.

AEs can be spontaneously reported or elicited during open-ended questioning, examination, or evaluation of a subject (in order to prevent reporting bias, subjects should not be questioned regarding the specific occurrence of one or more AEs).

Any AE must be reported by an entry in the eCRF within 5 days of awareness, even if they do not meet the whole information. The diagnosis of the event should be recorded as AE term. If there is a secondary AE separated in time from the initiating event, it should be recorded as an independent event (e.g., if vomiting results in severe dehydration, both events should be reported separately).

#### 13.2. Definition of Serious Adverse Event (SAE) and Suspected Unexpected



# **Serious Adverse Reaction (SUSAR)**

A Serious Adverse Event (SAE) is defined in general as any undesirable medical occurrence/adverse drug experience that occurs from the subject's written consent to participate in the study through **30** days after the final administration of the IMP, regardless of whether it is considered related or not to the study drug and that, at any dose, results in any of the following:

- results in death (fatal),
- is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it was more severe),
- requires inpatient hospitalization or causes prolongation of existing hospitalization (see NOTE 2 below),
- results in persistent or significant disability/incapacity,
- is a congenital anomaly/birth defect,
- is an important medical event. Defined as a medical event(s) that may not be immediately lifethreatening or result in death or hospitalization but, based upon appropriate medical and scientific judgment, may jeopardize the subject or may require intervention (e.g., medical, surgical, laboratory abnormal parameters...) to prevent one of the other serious outcomes listed in the definition above (see **NOTE 3** below),

After informed consent has been obtained, but prior to initiation of study drug, only serious adverse events caused by a protocol-mandated intervention (e.g., invasive procedures such as biopsies, discontinuation of medications) should be reported.

Seriousness is based on patient/event outcome or action criteria usually associated with events that pose a threat to a patient's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations

#### **NOTE 2**: The following hospitalizations are not considered SAEs:

- A visit to the emergency room or other hospital department < 24 hours, that does not result
  in admission, except if it is considered as an important medical event or life- threatening,</li>
- elective surgery, planned prior to signing consent,
- routine health assessment requiring admission for baseline/trending of health status (e.g., routine colonoscopy),
- admissions as per protocol for a planned medical/surgical procedure,
- admission for administration of anticancer therapy in the absence of any other SAEs,



- admission encountered for another life circumstance that carries no bearing on health status and requires no medical/surgical intervention (e.g., lack of housing, economic inadequacy, caregiver respite, family circumstances, administrative reason),
- progression of disease. By convention, clinical events related to the primary cancer being studied or to the primary cancer progression are not to be reported as SAEs, even if they meet any of the seriousness criteria from the standard SAE definition, unless the event is more severe than expected and therefore the investigator considers that their clinical significance deserves reporting.

**NOTE 3**: Any laboratory abnormalities should be documented as a SAE if:

- Intensive treatment in an emergency room or at home for allergic bronchospasm is needed,
- Blood dyscrasias or convulsions that do not result in hospitalization,
- Any untoward event related, and unexpected, to the protocol procedures,
- The laboratory test result is clinically significant or meets the definition of a SAE,
- The laboratory abnormality required the participant to have study drug discontinued or interrupted,
- The laboratory abnormality required the subject to receive specific corrective therapy.

A SAE report should be completed for any event where doubt exists regarding its seriousness. Although overdose, pregnancy, AESI (e.g., potential drug-induced liver injury (DILI)), important medical event, and cancer (secondary malignancy) are not always serious by regulatory definition, these events must be handled as SAEs. If applicable, SAEs must be collected that relate to any later protocol-specified procedure (e.g., a follow-up skin biopsy).

If the investigator believes that a SAE is not related to study drug but is potentially related to the conditions of the study (such as withdrawal of previous therapy or a complication of a study procedure), the relationship should be specified in the narrative section of the SAE Report Form and an important medical event would be the seriousness.

All deaths that occur during the reporting period that are clearly the result of disease progression should not be reported as a SAE, but they should be collected as an AE. All deaths where it is not due to disease progression and deaths with an unknown cause should always be reported as a SAE.

Death should be considered as an outcome and not the event, the AE causing the death must be reported as the SAE term. The term "sudden death" should be used only for the occurrence of an abrupt and unexpected death due to presumed cardiac causes in a patient with or without preexisting heart disease, within 1 hour after the onset of acute symptoms or, in the case of an unwitnessed death, within 24 hours after the patient was last seen alive and stable. If the cause of



death is unknown and cannot be ascertained at the time of reporting, "Death due to Unknown Cause" should be recorded on the Adverse Event eCRF. If the cause of death later becomes available (e.g., after autopsy), the event should be replaced by the established cause of death.

If the SAE is considered as related to the study drug by the Principal Investigator, it is a Serious Adverse Reaction. The SAR is assessed by the Fundación GECP (SLCG/GECP) to know if it is expected. A SAR that is not listed as a known toxicity of the investigational drug in the summary of product characteristics (Investigator Brochure or Data Sheet) will be considered as a Suspected Unexpected Serious Adverse Reaction (SUSAR). The sponsor will inform to the Principal Investigator that this SAE has been considered as a SUSAR. In Spain, Health authority (AEMPS: Agencia Española del Medicamento y Productos Sanitarios) will also be informed about all SUSARs via EudraVigilance. Also, the autonomous regions will be informed about all SUSARs according to the current Spanish clinical trial regulation.

# **13.3.** Adverse events of Special Interest for Atezolizumab (Immediately reportable to the Sponsor)









# 13.5. SAEs and SUSARs reporting

Anν

SAE must be reported by submitting the completed Initial SAE Form in the online eCRF within 24 hours of awareness, even if they do not meet any of the seriousness criteria.

In case of the eCRF is unavailability, the submission could be done by sending the SAE form preferably by email to

An appropriate SAE form (see appendix 3), should be used to report SAEs to Fundación GECP (SLCG/GECP). The paper SAE form has to be sent within the timeline period for reporting of 24 hours of awareness. **Once the eCRF system is available again, the SAE has to be completed and submitted by the site into the eCRF**.

If only limited information is initially available, a follow-up report is required to complete the information as soon as possible. (Note: Follow-up SAE reports should include the same SAE term(s) initially reported.)

The SAE outcome must be reported within 14 days after initial reporting by submitting the Follow up SAE Form in the online eCRF. In case the SAE is reported as ongoing after 14 days, a follow-up report has to be submitted again with the final outcome.

If an ongoing SAE changes in its grade, relationship to study drug, seriousness, SAE term or if new information becomes available, a new follow-up SAE report should be sent within 24 hours to the Fundación GECP (SLCG/GECP) using the same procedure after described.

Any SUSAR occurred during the trial will be notified under Spanish clinical regulation to the principal investigators, to the Health Authority (AEMPS) via Eudravigilance within the timelines specified in



the Royal Decree 1090/2015 on clinical trials regarding the recording, evaluation and reporting of adverse events. Also, the autonomous regions will be informed about all SUSARs according to the current Spanish clinical trial regulation.

For any doubt please contact Fundation GECP (SLCG/GECP) pharmacovigilance office by this email:

| Also, Fundación GECP (SLCG/GECP) will ensure that all SAEs, SUSARs, AESIs and pregnancy reports in the clinical database (eCRF) are reported to the authorization holder y during the conduct of the study including periodic reconciliation. |
|---|


# 13.7. Other safety considerations

Any significant worsening noted during interim or final physical examinations, electrocardiograms, X-rays, and any other potential safety assessments, whether or not these procedures are required by the protocol, should also be recorded as a non-serious or serious AE, as appropriate, and reported accordingly.

# 13.8. Adverse events related to the treatment and associated risks

| <u>ATEZOLIZUMAB</u> |
|---------------------|
| <u>BEVACIZUMAB</u> |





# 14. Biological material and translational research



 $<sup>{}^*\ \</sup>text{If the submitted tumor sample is insufficient or not valid to evaluate the TMB, a blood sample can be sent instead}\ .$ 



| _ | | |
|---|----|----------|
| | ı. | |
| | | <u> </u> |



# 15. Case report forms and documentation

eCRFs will only be available on-line at the Remote Data Entry (RDE) facility of Fundación GECP for patient enrollment.

Only the patient pre-screening form will be used in a paper form and will be send scanned by email or by fax (+34 93 419 17 68) to obtain the pre-screening number.

Also, another exception will be a paper SAE form and pregnancy form that will be used only in case of eCRF system unavailability.

#### 16. Statistical considerations

Three populations will be considered for different analyses:

• Per protocol population (PP): Per protocol population will consider patients that will receive a minimum of two cycles of atezolizumab and Bevacizumab or that have at least the first tumor response evaluation carried out. Patients without any radiological evaluation who may die during the first 12 weeks will also be considered PP population. Patients without the first tumor response evaluation carried out but with a progression disease (also clinical progression) at 6 weeks will also be considered into PP population.



- Intention to treat analysis (ITT): Intention to treat analysis will include all patients that will be registered into the clinical trial.
- Safety population (SFP): Safety population will include all patients that will be exposed to study treatment (atezolizumab + bevacizumab), whatever will be the quantity received

The primary endpoint is Progression Free Survival at 12 months (PFS) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

For one arm, we estimate to achieve a PFS at 12 months of 40% (vs 18% from Chemotherapy, previous published studies), with a 90% power and alpha 5%, one-sided test. The test statistic for survival probability is based on the non-parametric estimate of the survival distribution. Additionally, estimating a 10% of errors, withdrawals or others, it will be necessary to recruit 40 patients in order to get the study objectives.

If the withdrawals are higher than 5%, so that in order to reach the proposed sample size, if a patient initially enrolled in the study does not fulfil the inclusion criteria, they will be replaced by a new one subject that fulfil them, this replacement will ensure that the sample size will be the one calculated initially.

#### Data analysis and statistical methods

A descriptive analysis will be made of the variables calculating absolute and relative frequencies of qualitative variables and mean(standard deviation) or median (25 and 75 percentiles), minimum and maximum values for quantitative variables.

For the primary endpoint analysis, survivor function estimated by Kaplan-Meier method will be used, as well as the survival curves.. The 95% confidence interval will be estimated.

For the bivariate analysis, appropriate parametric and nonparametric tests will be used depending on whether the data are normally or non-normally distributed. For comparison of quantitative variables, Student's t test for independent data, the Mann-Whitney U test, analysis of variance or the Kruskal-Wallis H test will be used.

#### 17. Criteria for termination of the trial

#### 17.1. General criteria for termination of the trial

The trial may be discontinued early in parts or completely if the information on the product leads to doubt as to the benefit/risk ratio, by decision of Fundación GECP or Trial Steering Committee, or at the suggestion of the IDMC.



The trial can be terminated at any time if the authorization and approval to conduct the study is withdrawn by ethics committee or regulatory authority decision, insufficient accrual, emerging new data impacting the scientific value of the trial or on ethical grounds.

# 17.2. Discontinuation of protocol treatment and from the study for individual patients

Patients may be withdrawn from the protocol treatment and from the study in the following situations:

- Occurrence of unacceptable toxicities. Stopping protocol treatment is determined by medical judgment of the treating physician.
- Disease progression per investigator assessment according to RECIST v1.1 and loss of clinical benefit
- Symptomatic deterioration attributed to clinical disease progression
- Inter-current severe illnesses which would in the judgment of the investigator affect assessments of the clinical status to a significant degree and require discontinuation of protocol therapy
- Request by the patient. Patients have the right to refuse further trial treatment at any time during the trial. Such patients will remain in the trial and will be transferred to the follow-up phase.
- If a patient refuses to have follow-up examinations and tests needed to determine whether the treatment is safe and effective
- Protocol non-compliance or study termination by sponsor or site closure by the sponsor (poor protocol adherence, inaccurate or incomplete data recording...)
- Pregnancy
- Patient non-compliance, defined as a failure to comply with the protocol requirements as determined by the protocol

The decision for discontinuation of protocol treatment and the study of individual patients is taken by the treating physician based on his medical evaluation and taking into account the patient's individual situation.

Specific reasons for trial discontinuation where further collection of data is not allowed are: withdrawal of consent, patient lost to follow up, death.

All possible measures will be undertaken to maintain the investigation program and to continue the follow-up even if the treatment was prematurely concluded and/or if the patient did not attend the follow-up visits at the participating institution.



The primary reason for the treatment and study discontinuation should be documented on the appropriate eCRF.

# 18. Ethics aspects, regulatory approval, and Patient Informed Consent

The Investigator will ensure that this study is conducted in full conformance with the principles of the "Declaration of Helsinki" or with the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the individual. The study must fully adhere to the principles outlined in "Guideline for Good Clinical Practice" ICH6 Tripartite Guideline (January 1997) or local Spanish law if it affords greater protection to the patient. For studies conducted in the EU/EEA countries, the Investigator will ensure compliance with the EU Clinical Trial Directive (2001/20/EC).

# 18.1. Ethical Review Board/Ethics Committee/Health Authority

All protocols and the patient informed consent forms must have the approval of a properly constituted committee or committees responsible for approving clinical trials. The Ethic Committee decision must contain approval of the designated investigator, the protocol (identifying protocol title and version number), and of the patient informed consent.

The Ethic Committee written, signed approval letter/form must contain approval of the designated investigator, the protocol (identifying protocol title and version number), and of the patient informed consent.

Any modifications made to the protocol must be submitted to the appropriate Ethic Committee for information or approval in accordance with local procedures and regulatory requirements and to Health Authorities if required.

Once approved or acknowledged by the appropriate ERB/IRB and by the Health Authorities (if required), the investigator shall implement the protocol modifications.

If applicable, in addition to the approval of the Ethics Committee according to national legislation, the protocol, other protocol related documents including patient information and informed consent and other documents as required locally must be submitted to and be approved by the health authority.

#### 18.2. Informed consent

Both Informed consent (pre-screening IC and IC for the study) for each patient will be obtained prior to initiating any trial procedures in accordance with the "Patient Information and Informed Consent". Once signed and dated, a copy of the informed consent must be given to each patient and the original copy must be retained in the investigator's site file. The informed consent form must be available in the case of data audits.



The "Declaration of Helsinki" recommends that consent be obtained from each potential patient in biomedical research trials after the aims, methods, anticipated benefits, and potential hazards of the trial, and discomfort it may entail, are explained to the individual by the physician. The potential patient should also be informed of her/his right to not participate or to withdraw from the trial at any time. The patient should be told that material from her/his tumor and blood and serum samples will be stored and potentially used for additional studies not described in this protocol.

If the patient is in a dependent relationship to the physician or gives consent under duress, the informed consent should be obtained by an independent physician. It is preferable that the patient who gives the consent signs the form but if it is not possible or if the patient is legally incompetent (i.e., a minor, or mentally incompetent), informed consent must be obtained from the parent, legal guardian, or legal representative in accordance with the law of the country in which the trial is to take place.

By signing this protocol, the investigator agrees to conduct the trial in accordance with Good Clinical Practice and the "Declaration of Helsinki".

The template Patient Information Sheet and Informed Consent has been written according to ICH guidelines which state the Informed Consent should adhere to GCP and to the ethical principles that have origin in the "Declaration of Helsinki".

### 19. Governance and administrative issues

# 19.1. Study documentation

The investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented, including, but not limited to, the protocol, protocol amendments, Informed Consent Forms, and documentation of IRB/EC and governmental approval.

## 19.2. Protocol non-compliances/deviations

The investigator should document and explain any protocol non-compliances/deviations.

#### 19.3. Protocol amendment

Any protocol amendments will be prepared by the Sponsor. Protocol amendments will be submitted to the IRB/EC and to regulatory authorities in accordance with local regulatory requirements. Approval must be obtained from the IRB/EC and regulatory authorities (as locally required) before



implementation of any changes, except for changes necessary to eliminate an immediate hazard to patients or changes that involve logistical or administrative aspects only (e.g., change in Medical Monitor or contact information).

### 19.4. Final report

A final clinical trial report will be written and distributed to the Ethic committees and Health Authorities as required by applicable regulatory requirements.

### 19.5. Independent Data Monitoring Committee

The trial will be presented periodically for review to the Fundación GECP BICR (blinded independent central review).

#### 19.6. Publication

Authorship on the final manuscript or publications or provisional extracts will be decided in accordance with the Fundación GECP publication and authorship guidelines (SOP GECP: Política de publicaciones y auditorías).

None of the participants will present data to his centre in isolation from the rest of the results of the study and will need to seek approval from the sponsor.

### 19.7. Financial disclosure

Investigators will provide the sponsor with enough, accurate financial information in accordance with local regulations to allow the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate health authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

#### 19.8. Clinical trial insurance

Spanish legislation demands cover with a civil responsibility policy for subjects participating in a clinical trial. Fundación GECP will contract the appropriate liability insurance for this trial. Patients who suffer injuries due to the trial should report them immediately to their physician.

### 19.9. Quality assurance

Fundación GECP conducts trials according to the ICH Good Clinical Practice (GCP) guidelines. The Trial Data Manager reviews each eCRF as per monitoring plan schedule.

Fundación GECP will conduct periodic triggered visits to the participating sites to ensure proper trial conduct, verify compliance with GCP, and perform source data verification.



The Investigator should ensure that source documents are made available to appropriately qualified personnel from Fundación GECP, or to ethics committee and health authority inspectors after appropriate notification.

At regular intervals during the clinical trial, the centre will be contacted, through monitoring visits, letters or telephone calls, by a representative of the Monitoring Team to review study progress, investigator and patient compliance with clinical trial protocol requirements and any emergent problems. These monitoring visits will include but not be limited to review of the following aspects: patient informed consent, patient recruitment and follow-up, SAE documentation and reporting, AEs with pre-specified monitoring documentation and reporting, AE documentation, dispensing IMP, compliance with protocol, drug accountability, concomitant therapy use, quality of data and storage of blood and serum samples.

#### 19.10. Data protection

The samples and data collected will be coded to protect patient confidentiality. Each patient will have a pre-screening number at the pre-screening phase to identify the biological material and a unique identifier assigned by the eCRF of the study once enrolled. Sites are responsible to keep a patient log locally in order to be able to link the pre-screening number and the unique identifier to the record of the patient.

No identifiable / personal data will be stored in the trial database or the tissue repositories in the central laboratories.

Regulatory authorities and pertinent Ethics Committees (IRB/ERB) may have access to patient data on-site. Fundación GECP audit or monitoring personnel will also have access to such data on-site.

In Spain to ensure the patient confidentiality of data applies from the 25<sup>th</sup> of May 2018 the Reglamento (UE) 2016/679 del Parlamento europeo y del Consejo de 27 de abril de 2016 de Protección de Datos (RGPD).

### 19.11. Study monitoring team

The Fundación GECP will be responsible for monitoring the trial at Spanish sites.

The clinical monitor is obliged to rigorously follow the study. For this, the clinical monitor will regularly visit the study centers and the investigators as well as maintain necessary written and telephone communications.

The clinical monitor will assess the data collected in the acquisition forms and compare them with the original data of the clinical history and other original documents in conjunction with the study investigator.

The contact persons will be:



Fundación GECP CRA Meridiana 358, 6ª planta 08027 Barcelona Tel. 93 430 20 06 Fax. 93 419 17 68

Fundación GECP Lead CRA Meridiana 358, 6ª planta 08027 Barcelona Tel. 93 430 20 06 Fax. 93 419 17 68

#### 19.12. Record retention

The centre must retain all essential documents according to ICH GCP. This includes copies of the patient trial records, which are considered as source data, patient informed consent statement, laboratory printouts, drug inventory and destruction logs, and all other information collected during the trial. These documents are to be stored until at least 25 years after the termination of the trial.

In the event that the Principal Investigator retires or changes employment, custody of the records may be transferred to another competent person who will accept responsibility for those records. Written notice of such transfer must be given to the Fundación GECP and the local Ethics Committee at least 1 month in advance.





| <u> </u> | |
|-------------|-----|
| | ı ı |
| <del></del> | |
| | I |



| _ |
|---|









| | _ |
|---|---|
| _ | |



### **Appendices:**

- 1. Common Terminology criteria for Adverse Events (CTCAE)
- 2. RECIST criteria v1.1
- 3. SAE Form
- 4. Pregnancy Form
- 5. Health-related Quality of life questionnaire: EORTC C30 (QLQ-C30) and submodule LC13
- 6. System of classification for non-microcytic lung cancer (NSCLC) and definition of lymph node maps, 8<sup>th</sup> edition
- 7. Risks associated with Atezolizumab and guidelines for management of adverse events associated with Atezolizumab
- 8. Patients pre-screening form TELMA
- 9. Foundation one CDx Specimen Instructions
- 10. Foundation one Liquid technical sheet
- 11. Foundation one CDx technical sheet

**APPENDIX 1**. Common Terminology criteria for Adverse Events (CTCAE)

Version 5.0: November 27, 2017 is available from the internet at:

https://ctep.cancer.gov/protocolDevelopment/electronic applications/docs/ CTCAE v5 Quick Reference 8.5x11.pdf



#### APPENDIX 2. RECIST criteria v1.1

#### 1. Introduction

All included patients will be evaluated for response according to the revised Response Evaluation Criteria In Solid Tumors (RECIST version 1.1) [1]. This appendix defines all criteria applied in this trial.

#### 2. Methods of assessment

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during follow-up. Imaging-based evaluation is preferred to evaluation by clinical examination when both methods have been used to assess the antitumor effect of a treatment.

**CT** is the best currently available and reproducible method to measure lesions selected for response assessment. CT should generally be performed using  $a \le 5$  mm contiguous reconstruction algorithm. **MRI** is acceptable for certain situations, e.g. body scans.

Clinical lesions will only be considered measurable when they are superficial (e.g. skin nodules) and ≥10 mm. In the case of skin lesions, documentation by color photography including a ruler to estimate the size of the lesion is recommended.

Lesions on **chest X-ray** are acceptable as measurable lesions when they are clearly defined and surrounded by aerated lung. However, CT is preferable.

**Ultrasound** is not useful in assessment of lesion size and is not accepted as method of assessment.

**FDG-PET** is not foreseen for regular response assessments. It may, however, be used to detect or confirm the appearance of new lesions. Attenuation correction CT scans performed as part of a **PET/CT** scan frequently show lower resolution; therefore, dedicated CT scans are preferred. However, if the site can demonstrate that the CT performed as part of a PET/CT is of the same diagnostic quality as a diagnostic CT (with IV and oral contrast), then the CT portion of the PET/CT can be used for RECIST measurements.

### 3. Measurability of tumor at baseline

Measurable disease is defined as the presence of at least one measurable lesion.

#### Measurable lesions:

- **Tumor lesions** must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of
  - o 10 mm by CT scan (CT scan slice thickness no greater than 5mm)



- 10mm caliper measurement by clinical exam (lesions which cannot be accurately measured with calipers should be recorded as non-measurable)
- o 20 mm by chest X-ray
- Malignant lymph nodes: to be considered pathologically enlarged and measurable, a lymph node must be ≥ 15mm in *short* axis when assessed by CT scan, assuming the slice thickness is ≤ 5 mm. At baseline and in follow-up, only the *short* axis will be measured.

#### Non-measurable lesions: all other lesions, i.e.:

- Small non-nodal lesions (longest diameter < 10 mm in CT scan)</li>
- Small lymph nodes (short axis ≥ 10 and < 15 mm). Lymph nodes that have a short axis < 10 mm are considered non-pathological and should not be recorded or followedBone lesions. Lytic bone lesions or mixed lytic-blastic lesions, with identifiable soft tissue components, can be considered as measurable lesions if the soft tissue component meets the definition of measurability described above. Blastic bone lesions are non-measurable.</p>
- Leptomeningeal disease
- Ascites
- Pleural or pericardial effusion
- Inflammatory breast disease
- Lymphangitic involvement of skin or lung
- Cystic lesions. Cystic lesions thought to represent cystic metastases may be considered as measurable lesions. However, if non-cystic lesions are present, these are preferred as target lesions
- Tumor lesions situated in a previously irradiated area, or subjected to other locoregional therapy. Such lesions may be considered measurable if there has been demonstrated progression in the lesion
- abdominal masses/abdominal organomegaly identified by physical exam that are not measurable by reproducible imaging techniques

#### 4. Selection of lesions

# 4.1. Selection of target lesions

At baseline, measurable lesions up to a maximum of 5 lesions representative of all involved organs, and up to 2 per organ, should be identified as target lesions and measured and recorded. Target lesions (TL) should be selected on the basis of their size and their suitability for accurate repetitive measurements. A sum of diameters for all target lesions will be calculated and reported as the baseline sum of diameters. Lymph nodes selected as TL should always have the short axis recorded. All other lesions should always have their longest diameters recorded. The sum of diameters will be used as reference to further characterize the objective tumor response of the measurable dimension of the disease.



#### 4.2. Selection of non-target lesions

All other lesions (or sites of disease) should be identified as non-target lesions and should also be recorded at baseline. Measurements are not required, but the presence or absence of each should be noted throughout follow-up. It is possible to record multiple non-target lesions as a single item on the CRF (e.g. "multiple liver metastases").

#### 5. Evaluation of Lesions

#### 5.1. Evaluation of Target Lesions

All target lesions will be measured at each tumor assessment, and the sum of their diameters will be compared to previous assessments in order to assign the response status as specified below.

- Complete Response (CR): Disappearance of all target lesions. Lymph nodes selected as target
  lesions must each have reduction in the short axis to < 10 mm in order for the response to
  be considered complete. In this case, the sum of diameters may be > 0.
- Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters.
- Progression (PD): At least a 20% increase in the sum of diameters of target lesions, taking as
  reference the smallest sum recorded on study. In addition to the relative increase of 20%,
  the sum must also demonstrate an absolute increase of at least 5 mm.
- Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum of diameters recorded on study.
- Inevaluable for response: specify reasons (for example: early death due to malignant disease or toxicity; tumor assessment not repeated/incomplete; other, specify).

**Note:** All target lesions, including lymph nodes, should have their actual measurements recorded at each subsequent evaluation, even when very small (e.g. 2 mm). If the radiologist does not feel comfortable assigning an exact measure and reports a lesion as "too small to measure", a default value of 5 mm should be recorded. If a TL is thought likely to have disappeared, "0 mm" is noted.

#### 5.2. Evaluation of Non-Target Lesions

- Complete Response (CR): Disappearance of all non-target lesions; lymph nodes selected as non-target lesions must be non-pathological in size (< 10 mm).
- Non-CR/non-PD: Persistence of one or more non-target lesions (non-CR).
- Progression (PD): unequivocal progression of existing non-target lesions. Unequivocal
  means: comparable in magnitude to the increase that would be required to declare PD for
  measurable disease, or an overall substantial increase in tumor burden that merits treatment
  discontinuation.



#### 5.3. Determination of new lesions

The appearance of any new malignant lesions denotes disease progression. The finding of a new lesion should be unequivocal, i.e. not attributable to differences in scanning technique or findings thought to represent something other than tumor. If a new lesion is equivocal, e.g. because of its small size, the patient will stay on treatment (if the decision on PD is based on this lesion only). If the repeat scans confirm there is definitely a new lesion, then progression should be declared using the date of the previous scan.

Lesions found in a new location not included in the baseline scan (e.g. brain metastases) are considered new lesions.

**Note:** the "re-appearance" of a previously "disappeared" target or non-target lesion does not in itself necessarily qualify as PD; this is the case only if the overall evaluation meets the PD criteria, or if the patient was previously in CR.

#### 5.4. Additional considerations

In some circumstances, it may be difficult to distinguish residual disease from normal tissue. When the evaluation of complete response depends upon this determination, it is recommended that the residual lesion be investigated (fine needle aspirate/biopsy) before confirming the complete response status.

The cytological confirmation of the neoplastic origin of any effusion that appears or worsens during treatment when the measurable tumor has met criteria for response or stable disease is mandatory to differentiate between response or stable disease (an effusion may be a side effect of the treatment) and progressive disease.

## 6. Determination of time point response

Based on the responses of Target Lesions, Non-Target Lesions, and the presence or absence of new lesions, the overall response will be determined at each tumor assessment time point, according to the table below:

| Target lesions | Non-target lesions | New lesions | Overall response |
|---|---|---|---|
| CR | CR | No | CR |
| CR | Non-CR / non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not all evaluated | No | PR |



| SD | Non-PD or not all evaluated | No | SD |
|---|---|---|---|
| Not all evaluated | Non-PD | No | NE<br>(unless the sum of<br>diam. Of evaluated<br>lesions indicates PD <sup>1</sup> ) |
| PD | Any | Yes or no | PD |
| Any | PD | Yes or no | PD |
| Any | Any | Yes | PD |

<sup>&</sup>lt;sup>1</sup> From ref. 1 p.234: When no imaging/measurement is done at all at a particular time point, the patient is not evaluable (NE) at that time point. If only a subset of lesion measurements are made at an assessment, usually the case is also considered NE at that time point, unless a convincing argument can be made that the contribution of the individual missing lesion(s) would not change the assigned time point response. This would be most likely to happen in the case of PD. For example, if a patient had a baseline sum of 50mm with three measured lesions and at follow-up only two lesions were assessed, but those gave a sum of 80 mm, the patient will have achieved PD status, regardless of the contribution of the missing lesion.

#### 7. Determination of best overall response

Best overall response is defined as best response across all time points. Confirmation of partial or complete response by an additional scan is not requested in this trial. Best overall response will be determined by central review.



# **APPENDIX 3**. SAE Form

| SERIOUS ADVERSE EVEN | TS NOTIFIC | CATION FORM (SAE) | Charles 1990 | OCOL Code: GECP<br>code: ML40237 | 18/03 (TELMA) | |
|---|---|---|---|---|---|---|
| Ge | CP | | Site: | | | |
| TYPE OF NOTIFICATION: | JP n <sup>R</sup> | | Invest | igator: | | SAE Form<br>Nr: |
| SERIOUS ADVERSE EVENT I | NFORMAT | ION | | | | , |
| PATIENT CODE | DAT | TE OF BIRTH | AGE | GENDER | WEIGHT (kg | HEIGHT (cm) |
| DATE OF SAE AWARENESS | : [] | | SAE NO | OTIFICATION DATE | E; II_ | 1 |
| SERIOUS ADVERSE EVENT<br>events. The first one has t<br>term according to the CTC<br>base. | o be the m | ore relevant. The SAE | term ha | is to be filled in w | ith the verbation | n term. The SAE |
| SAE term | Grade<br>(1-5) | Start Date/Stop | date | Causality <sup>1</sup> | Key for seriousness <sup>2</sup> | Outcome <sup>3</sup> |
| | | Start D.: III | t | | | |
| S7 | es e | Stop D.: III | _1 | • | | Outcome date: |
| | | Start D.: III_ | | | | |
| | | Stop D.: III_ | _1 | • | | |
| | | Start D.: III | | | | |
| 97 | | Stop D.: III_ | _1 | • | | |
| | | Start D.: III_ | | 20 | į. | |
| 3 | es - s | Stop D.: III_ | _1 | • | | |
| | | Start D.: III_ | | 1 | ć. | |
| 3 | | Stop D.: III | _1 | | | |
| <sup>1</sup> Causality (relation to study | drugs): | ² Key for | r Seriousn | iess: | 3 Ou | tcome |
| O: Not related; 1: Related*; 2<br>applicable<br>*Specify drug and/or therapy<br>Radiotherapy) | | 1: Death; 2: Life threat<br>hospitalization admiss<br>Anomaly/Birth Defect<br>Disability; 6: Medical<br>medical event); 7: No<br>special interest (AESI)<br>serious secondary mai | sion; 4:Co<br>;5: Persist<br>lly signific<br>on-serious<br>as per pro | ngenital<br>tent or significant<br>ant (important<br>adverse event of<br>otocol; 8: Non- | 196. TA 2700 Lab (1962) (1962) | hout sequelae ; 2:<br>equelae; 3: Fatal;<br>nknown |
| SAE COMMENTS (Please, poi<br>of death, please add informat | The second second second | | | A SEC AND SERVICE | tional relevant in | formation, in case |

Protocol\_

SAE Form\_v.5.0\_16Abr2019



| PATIENT CODE | | GECP 18/0 | | COL CODE<br>_Roche code: M | L40237 | SAE FORM N' | |
|---|---|---|---|---|---|---|---|
| NFORMATION ABOUT IN | IVESTIGATI | ONAL MEDI | CAL PROD | OUCT | | | |
| Trial Medication<br>(Generic name/Brand<br>name) | Dose and u | Rout<br>(IV, P<br>SC | O, Date | of administration<br>before SAE | Action<br>taken <sup>4</sup> | Stopped the<br>event when the<br>medication was<br>discontinued? <sup>5</sup> | The event returne<br>when the<br>medication is<br>resumed? <sup>5</sup> |
| | | | 3 | | | | |
| AIS THERE ANY OTHER EXPLANATION | | | | TUDY PROCEDURES | NOT APPLICABLE | E ☐ OTHERS (SPECIFY): | 3: |
| Action taken with regard<br>discontinuation; 5: other (s<br>Stopped or returned the a<br>REVIOUS RELEVANT ME | pecify):<br>idverse even | it when the n | | | | | |
| PREVIOUS RELEVANT MEDICAL HI | | 2307 | URGERIES, A | LLERGY, PREGNANCI | ES, CONCOMITA | ANT DISEASES, ETC): | |
| ONCOMITANT MEDICAT CONCOMITANT MEDIC (Brand name) | 1// | Daily Dose | Route<br>(IV, PO,<br>SC) | basal diseases or su<br>Onset Date | eportive Clinica<br>Ending dat<br>Ongoing | te or Preso | ription reason <sup>6</sup> |
| | | | ** | | | | |
| Prescription reason: 1: Regul | ar medication | ı/baseline con | ditions: 2: 0 | oncomitant Medi | cation/proph | vlaxis: 3: Adverse ev | ent: 4: Other |
| specify)<br>NFORMATION ABOUT TH | | d : Se. S | 200-1, N2:0418 | de hit breed to the material | 1000124-0476-0411 | | 194511. 090611. |
| NAME AND CONTACT DETAILS OF THE SPONSOR Fundación GECP Av. Meridiana, 358 6º pl 08027 Barcelona Tel: (34) 93 430 20 06 Fax: (34) 93 419 17 68 | Section and the | EIVED AND S | | egymnoren erest<br>e Banaevereste | ONTACT | Pagadonas | IGNATURE OF |

SAE Form\_v.5.0\_16Abr2019



# **APPENDIX 4**. Pregnancy Form

| PREGNANCY NOTIFICA | ATION FORM | | OCOL Code: GECP 18<br>code: ML40237 | 3/03 (TELI | MA) | |
|---|---|---|---|---|---|---|
| Gec | P | Site: | | | | |
| TYPE OF NOTIFICATION: □ INITIAL □ FOLLOW UP n <sup>R</sup> | | Invest | igator: | | 200 | SNANCY<br>n Nr: |
| PATIENT CODE I | DATE OF BIRTH | AGE | GENDER | WEIGHT | T (kg) | HEIGHT (cm) |
| DATE OF PREGNANCY AWARENES | S: III | I PREG | NANCY NOTIF. DAT | E: I | 1 | |
| PREGNANCY REPORT INFORMATION | ON | | | | | |
| *If in pregnant trial subject. Was sh<br>** Date of withdrawal of the study<br>State of the pregnancy at the mome | <u> </u> | 11 | | ty test 🗆 | Confin | med |
| PHASE OF THE TREATMENT WHEF | RE PREGNANCY WA | S DETECTED A | IND TYPE OF CLINICA | AL TRIAL | | |
| □ Screening Phase □ Randomized<br>Is it a blind Clinical trial? □ NO □ | 170 | 1,500 | 17.0 | s* | | |
| \ <del>-</del> | 170 | s the blind brok | sen? □ NO □ YE | 1 | 200 | |
| Is it a blind Clinical trial? *Specify (treatment arm, treatment): MATERNAL INFORMATION Mother date of birth: | 170 | s the blind brok | 17.0 | ation: | metho | |
| Is it a blind Clinical trial? NO Specify (treatment arm, treatment): MATERNAL INFORMATION Mother date of birth: Date of last menstrual period: | 170 | s the blind brok | ntraception informations the mother/fathentraception? | ation:<br>r using a | | |
| Is it a blind Clinical trial? *Specify (treatment arm, treatment): MATERNAL INFORMATION Mother date of birth: | 170 | I Co | ntraception informations the mother/fathentraception? | ation: r using a es* coception | □ No | od of |
| Is it a blind Clinical trial? NO Specify (treatment arm, treatment): MATERNAL INFORMATION Mother date of birth: Date of last menstrual period: Estimated delivery date: | 170 | I Co | en? D NO D YE Intraception informations the mother/father intraception? D You pecify: D Oral contral | ation: r using a es* proception s (specify | □ No<br>□ Con | od of<br>ndom |
| Is it a blind Clinical trial? *Specify (treatment arm, treatment): MATERNAL INFORMATION Mother date of birth: Date of last menstrual period: Estimated delivery date: Father date of birth: | YES; If yes, Wa | I Co | en? DNO PE | ation: r using a es* c sception s (specify evious pr | □ No<br>□ Con<br>():<br>regnan | od of odom |
| Is it a blind Clinical trial? *Specify (treatment arm, treatment): MATERNAL INFORMATION Mother date of birth: Date of last menstrual period: Estimated delivery date: Father date of birth: First pregnancy awareness date: | YES; If yes, War | I Co | ntraception informations as the mother/fathentraception? Your pecify: Oral contraction program Otherwise the mother any program of the program Otherwise the mother any program Oral program Otherwise the mother any program Oral program Otherwise the mother any program Otherwise the mother any program Oral program Otherwise the mother any program Oral program Oral program | ation: r using a es* c sception s (specify evious pr | □ No<br>□ Con<br>():<br>regnan | od of odom |
| Is it a blind Clinical trial? *Specify (treatment arm, treatment): MATERNAL INFORMATION Mother date of birth: Date of last menstrual period: Estimated delivery date: Father date of birth: First pregnancy awareness date: PI awareness date of the pregnance | I YES; If yes, Was | I Co | ntraception informations as the mother/fathentraception? Your pecify: Oral contraction program Otherwise the mother any program of the program Otherwise the mother any program Oral program Otherwise the mother any program Oral program Otherwise the mother any program Otherwise the mother any program Oral program Otherwise the mother any program Oral program Oral program | ation: r using a es* c acception s (specify evious pr section) | □ No<br>□ Con<br>():<br>regnan | od of indom |
| Is it a blind Clinical trial? *Specify (treatment arm, treatment): MATERNAL INFORMATION Mother date of birth: Date of last menstrual period: Estimated delivery date: Father date of birth: First pregnancy awareness date: PI awareness date of the pregnance of the preg | YES; If yes, Was | the blind broken in the bl | ntraception informates the mother/fathentraception? | ation: r using a es* : eception s (specify evious pr section) | □ No<br>□ Con<br>():<br>regnan | od of odom |

Pregnancy Notification Form\_v.3.0\_26Abr2019

2 de 3



| PATIENT CODE | | PROTOCOL CODE GECP 18/03 (TELMA)_Roche code: ML40237 | | | L40237 | PREGNANCY Form N' | |
|---|---|---|---|---|---|---|---|
| REVIOUS RELEVANT MEDICAL | HISTORY FF | ROM MOT | HER AND | OR FATH | ER | | |
| PREVIOUS RELEVANT MEDICAL HISTORY ( | PREVIOUS DIAGNO | SIS, SURGERIES, | ALLERGY, CON | COMITANT DISE | EASES, ETC): | | |
| NFORMATION ABOUT INVEST | IGATIONAL I | MEDICAL F | | | - | | |
| Trial medication<br>(Generic name/Brand name) | Time of exposure! | Daily<br>dose | Route<br>(IV, PO,<br>SC) | Start D | ate | p date or<br>ngoing? | Action taken with rega<br>to trial medication <sup>2</sup> |
| Time of exposure: 0: pre-concep<br>Action taken with regard to tria<br>I: permanent discontinuation; 5:<br>ONCOMITANT MEDICATION ( | l medication:<br>other (specif | 0: None; 1<br>y): | : Reduced | ; 2: Delayed | d; 3: Delayed a | 100 1440 | no Car oso rom |
| CONCOMITANT MEDICATION<br>(Brand name) | - 8 | Rou | ite<br>PO, On | set Date | Ending date<br>Ongoing? | or | Prescription reason <sup>3</sup> |
| | | * | | | \$ | 28 | |
| | | | | | <u> </u> | 31 | |
| Prescription reason: 1: Regular of the properties of the propertie | medication/b | aseline con | ditions; 2 | Concomit | ant medicatio | n/prophyla | xis; 3: Adverse Event; |
| CURRENT PREGNANCY STATUS | AND OUTC | OME | | | | | |
| ONGOING - Yes - No (com | nplete sectio | n) = Hoke | | 500 BBS 0 | Varia 87 A | 98 | |
| □ Lost to follow u | | | | Newborn<br>(delivery | | | |
| □ Lost to follow u | | | | (delivery | date)<br>mode: □ vag | | arian |
| □ Lost to follow u | | | | (delivery<br>Delivery r | date)<br>mode: □ vag | inal 🗆 caes<br>known/oth | arian<br>ners: |
| | p: II_ | | 1 | (delivery r<br>Delivery r<br>Gestation | date)<br>mode: □ vag<br>□ Uni<br>al weeks at l | inal = caes<br>known/oth<br>pirth: I | arian<br>ners: |
| Lost to follow under the lost to follow under | p: II_ | | | (delivery r<br>Delivery r<br>Gestation<br>Duration | date)<br>mode: □ vag<br>□ Uni<br>al weeks at l | inal = caes<br>known/oth<br>birth: lhou | arian ners:I ursminutes |

Pregnancy Notification Form\_v.3.0\_26Abr2019



| PATIENT CODE | - TO | | DCOL CODE<br>A)_Roche code: ML40237 | | PREGNANCY Form N° |
|---|---|---|---|---|---|
| IEWBORN BABY INFORM | | ach enfant) | | | |
| Number of babies: I | J | | Gender: Mai | e 🗆 Female | |
| Apgar 1 min5 | min | _10 min | Weight (Kg): | Height (cm): | Head circumference (cm): |
| If any abnormality in the newborn appeared, then answer the following question: Are there any hints that these incidences may be related to the drug exposure of the mother/father during pregnancy? YES (complete SAE Form) | | | General status | of the newb | orn baby (specify): |
| VEORMATION ABOUT TH | IF STAFE W | I'HO ATTENDED THE | DELIVERY | | |
| | IE STAFF W | PEDIATRICIAN: | DELIVERY | ОТНЕЯ | ns: |
| NFORMATION ABOUT TH<br>GYNECOLOGIST:<br>NFORMATION ABOUT TH | | PEDIATRICIAN: | | | 0.453000 |
| GYNECOLOGIST: | IE SPONSO | PEDIATRICIAN: R AND THE PRINCI EIVED AND SIGNATU PONSOR: | PAL INVESTIGATO | OR (PI) OF TH | DATE AND SIGNATURE OF<br>THE PI: |
| GYNECOLOGIST: NFORMATION ABOUT TH IAME AND CONTACT PETAILS OF THE SPONSOR Fundación GECP Av. Meridiana, 358 6º pl 08027 Barcelona Tel: (34) 93 430 20 06 Fax: (34) 93 419 17 68 | DATE RECOFTHE SE | PEDIATRICIAN: R AND THE PRINCIPONSOR: | PAL INVESTIGATO | OR (PI) OF THE | E TRIAL DATE AND SIGNATURE OF |

3 de 3

Pregnancy Notification Form\_v.3.0\_26Abr2019



# APPENDIX 5. Health-related Quality of life questionnaire: EORTC C30 (QLQ-C30) and submodule LC13

Please see documents attached to the protocol

# APPENDIX 6. System of classification for non-microcytic lung cancer (NSCLC) and definition of lymph node maps, 8th edition

| T: Primary tumor | |
|---|---|
| Tx | Primary tumor cannot be assessed or tumor proven by presence of malignant cells in sputum<br>or bronchial washings but not visualized by imaging or bronchoscopy |
| TO TO | No evidence of primary tumor |
| Tis | Carcinoma in situ |
| T1 | Tumor $\leq$ 3 cm in greatest dimension surrounded by lung or visceral pleura without bronchoscopic evidence of invasion more proximal than the lobar bronchus (i.e., not in the main bronchus) <sup>a</sup> |
| T1a(mi) | Minimally invasive adenocarcinoma |
| T1a | Tumor ≤1 cm in greatest dimension |
| T1b | Tumor >1 cm but ≤2 cm in greatest dimension* |
| T1c | Tumor >2 cm but ≤3 cm in greatest dimension® |
| T2 | Tumor $>$ 3 cm but $\leq$ 5 cm or tumor with any of the following features <sup>c</sup> : |
| | <ul> <li>Involves main bronchus regardless of distance from the carina but without involvement<br/>of the carina</li> </ul> |
| | - Invades visceral pleura |
| | <ul> <li>Associated with atelectasis or obstructive pneumonitis that extends to the hilar region,<br/>involving part or all of the lung</li> </ul> |
| T2a | Tumor >3 cm but ≤4 cm in greatest dimension |
| T2b | Tumor >4 cm but ≤5 cm in greatest dimension |
| тз | Tumor >5 cm but ≤7 cm in greatest dimension or associated with separate tumor nodule(s) in the same lobe as the primary tumor or directly invades any of the following structures: chest wall (including the parietal pleura and superior sulcus tumors), phrenic nerve, parietal pericardium |
| T4 | Tumor >7 cm in greatest dimension or associated with separate tumor nodule(s) in a different<br>ipsilateral lobe than that of the primary tumor or invades any of the following structures:<br>diaphragm, mediastinum, heart, great vessels, trachea, recurrent laryngeal nerve, esophagus<br>vertebral body, and carina |
| N: Regional lymph node in | volvement |
| Nx | Regional lymph nodes cannot be assessed |
| NO NO | No regional lymph node metastasis |
| N1 | Metastasis in ipsilateral peribronchial and/or ipsilateral hilar lymph nodes and intrapulmonary<br>nodes, including involvement by direct extension |
| N2 | Metastasis in ipsilateral mediastinal and/or subcarinal lymph node(s) |
| N3 | Metastasis in contralateral mediastinal, contralateral hilar, ipsilateral or contralateral scalene,<br>or supraclavicular lymph node(s) |
| M: Distant metastasis | |
| MO | No distant metastasis |
| M1 | Distant metastasis present |
| M1a | Separate tumor nodule(s) in a contralateral lobe; tumor with pleural or pericardial nodule(s) or malignant pleural or pericardial effusion <sup>d</sup> |
| M1b | Single extrathoracic metastasise |
| M1c | Multiple extrathoracic metastases in one or more organs |

proximal to the main bronchus, is also classified as T1a.

Solitary adenocarcinoma,  $\leq$  3cm with a predominately lepidic pattern and  $\leq$  5mm invasion in any one focus. TZ tumors with these features are classified as TZa if  $\leq$ 4 cm in greatest dimension or if size cannot be determined, and TZb if >4 cm but

<sup>25</sup> cm in greatest dimension.

Most pleural (pericardial) effusions with lung cancer are due to tumor. In a few patients, however, multiple microscopic examinations of pleural (pericardial) fluid are negative for tumor and the fluid is nonbloody and not an exudate. When these elements and clinical judgment dictate that the effusion is not related to the tumor, the effusion should be excluded as a staging descriptor.

This includes involvement of a single distant (nonregional) lymph node.



| Occult carcinoma | TX | NO | MO |
|------------------|-----------|-----------|------------|
| Stage 0 | Tis | NO | MO |
| Stage IA1 | T1(mi) | NO | MO |
| | T1a | NO | MO |
| Stage IA2 | T1b | NO | MO |
| Stage IA3 | T1c | NO NO | MO |
| Stage IB | T2a | NO | MO |
| Stage IIA | T2b | NO NO | MO |
| Stage IIB | T1a-c | <u>N1</u> | MO |
| | T2a | N1 | MO |
| | T2b | N1 | MO |
| | T3 | NO | MO |
| Stage IIIA | T1a-c | N2 | MO |
| | T2a-b | N2 | MO |
| | T3 | N1 | MO |
| | T4 | NO | MO |
| | T4 | N1 | MO |
| Stage IIIB | T1a-c | <u>N3</u> | MO |
| | T2a-b | N3 | MO |
| | <u>T3</u> | N2 | MO |
| | T4 | N2 | MO |
| Stage IIIC | <u>T3</u> | <u>N3</u> | MO |
| | <u>T4</u> | N3 | MO |
| Stage IVA | Any T | Any N | M1a |
| | Any T | Any N | M1b |
| Stage IVB | Any T | Any N | <u>M1c</u> |



# **APPENDIX 7.** Risks associated with Atezolizumab and guidelines for management of adverse events associated with Atezolizumab

Toxicities associated or possibly associated with atezolizumab treatment should be managed according to standard medical practice. Additional tests, such as autoimmune serology or biopsies, should be used to evaluate for a possible immunogenic etiology, when clinically indicated.

Although most immune-mediated adverse events observed with immunomodulatory agents have been mild and self-limiting, such events should be recognized early and treated promptly to avoid potential major complications. Discontinuation of atezolizumab may not have an immediate therapeutic effect, and in severe cases, immune-mediated toxicities may require acute management with topical corticosteroids, systemic corticosteroids, or other immunosuppressive agents.

The investigator should consider the benefit-risk balance a given patient may be experiencing prior to further administration of atezolizumab. In patients who have met the criteria for permanent discontinuation, resumption of atezolizumab may be considered if the patient is deriving benefit and has fully recovered from the immune-mediated event. The decision to rechallenge patients with atezolizumab should be based on investigator's assessment of benefit-risk and documented by the investigator (or an appropriate delegate). Medical Monitor is available to advise as needed. Guidelines for managing patients who experience selected adverse events are provided in the following sections. Management guidelines are presented by adverse event severity based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE).

#### **PULMONARY EVENTS**

Dyspnea, cough, fatigue, hypoxia, pneumonitis, and pulmonary infiltrates have been associated with the administration of atezolizumab. Patients will be assessed for pulmonary signs and symptoms throughout the study and will have computed tomography (CT) scans of the chest performed at every tumor assessment.

All pulmonary events should be thoroughly evaluated for other commonly reported etiologies such as pneumonia or other infection, lymphangitic carcinomatosis, pulmonary embolism, heart failure, chronic obstructive pulmonary disease, or pulmonary hypertension. Management guidelines for pulmonary events are provided in Table 1.



**Table 1 Management Guidelines for Pulmonary Events, Including Pneumonitis** 

| Event | Management |
|---|---|
| Pulmonary<br>event, Grade 1 | Continue atezolizumab and monitor closely. Re-evaluate on serial imaging. Consider patient referral to pulmonary specialist. For Grade 1 pneumonitis, consider withholding atezolizumab |
| Pulmonary<br>event, Grade 2 | <ul> <li>Withhold atezolizumab for up to 12 weeks after event onset. <sup>a</sup></li> <li>Refer patient to pulmonary and infectious disease specialists and consider bronchoscopy or BAL.</li> <li>Initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day oral prednisone.</li> <li>If event resolves to Grade 1 or better, resume atezolizumab. <sup>b</sup></li> <li>If event does not resolve to Grade 1 or better while withholding atezolizumab, permanently discontinue atezolizumab and contact Medical Monitor. <sup>c</sup></li> <li>For recurrent events or events with no improvement after 48–72 hours of corticosteroids, treat as a Grade 3 or 4 event.</li> </ul> |
| Pulmonary<br>event, Grade 3<br>or 4 | <ul> <li>Permanently discontinue atezolizumab and contact Medical Monitor. ○</li> <li>Bronchoscopy or BAL is recommended.</li> <li>Initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day IV methylprednisolone.</li> <li>If event does not improve within 48 hours after initiating corticosteroids, consider adding an immunosuppressive agent.</li> <li>If event resolves to Grade 1 or better, taper corticosteroids over ≥1 month.</li> </ul> |

BAL=bronchoscopic alveolar lavage.

- <sup>a</sup> Atezolizumab may be withheld for a longer period of time (i.e., >12 weeks after event onset) to allow for corticosteroids (if initiated) to be reduced to the equivalent of ≤10 mg/day oral prednisone. The acceptable length of the extended period of time must be based on assessment of benefit-risk by the investigator and in alignment with the protocol requirement for duration of treatment and documented by the investigator. Medical Monitor is available to advise as needed.
- b If corticosteroids have been initiated, they must be tapered over ≥1 month to the equivalent of ≤10 mg/day oral prednisone before atezolizumab can be resumed.
- c Resumption of atezolizumab may be considered in patients who are deriving benefit and have fully recovered from the immune-mediated event. The decision to rechallenge patients with atezolizumab should be based on investigator's assessment of benefit-risk and documented by the investigator (or an appropriate delegate). Medical Monitor is available to advise as needed.

#### **HEPATIC EVENTS**

Immune-mediated hepatitis has been associated with the administration of atezolizumab. Eligible patients must have adequate liver function, as manifested by measurements of total bilirubin and hepatic transaminases, and liver function will be monitored throughout study treatment. Management guidelines for hepatic events are provided in Table 2.



Patients with right upper-quadrant abdominal pain and/or unexplained nausea or vomiting should have liver function tests (LFTs) performed immediately and reviewed before administration of the next dose of study drug.

For patients with elevated LFTs, concurrent medication, viral hepatitis, and toxic or neoplastic etiologies should be considered and addressed, as appropriate.

**Table 2 Management Guidelines for Hepatic Events** 

| Event | Management |
|---|---|
| In patients withou | ut HCC |
| Hepatic event,<br>Grade 1 | <ul> <li>Continue atezolizumab.</li> <li>Monitor LFTs until values resolve to within normal limits or to baseline values.</li> </ul> |
| Hepatic event,<br>Grade 2 | All events: Monitor LFTs more frequently until return to baseline values. Events of > 5 days' duration: Withhold atezolizumab for up to 12 weeks after event onset. Initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day oral prednisone. If event resolves to Grade 1 or better, resume atezolizumab. If event does not resolve to Grade 1 or better while withholding atezolizumab, permanently discontinue atezolizumab and contact Medical Monitor. **Open Company Com |
| Hepatic event,<br>Grade 3 or 4 | <ul> <li>Permanently discontinue atezolizumab and contact Medical Monitor. <sup>c</sup></li> <li>Consider patient referral to GI specialist for evaluation and liver biopsy to establish etiology of hepatic injury.</li> <li>Initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day oral prednisone.</li> <li>If event does not improve within 48 hours after initiating corticosteroids, consider adding an immunosuppressive agent.</li> <li>If event resolves to Grade 1 or better, taper corticosteroids over ≥ 1 month.</li> </ul> |



| Event | Management |
|---|---|
| In patients with HCC | |
| AST/ALT is within normal<br>limits at baseline and<br>increases to<br>>3×ULN to ≤10×ULN | Monitor LFTs more frequently until return to baseline values. Withhold atezolizumab for up to 12 weeks after event onset. |
| | Events of > 5 days' duration: |
| or | <ul> <li>Consider initiating treatment with corticosteroids equivalent to<br/>1–2 mg/kg/day oral prednisone.</li> </ul> |
| AST/ALT is >ULN to<br>≤3×ULN at baseline and | <ul> <li>If event resolves to baseline or to Grade 1 or better, resume<br/>atezolizumab.</li> </ul> |
| increases to<br>>5×ULN to ≤10×ULN | <ul> <li>If event does not resolve to baseline or to Grade 1 or better<br/>while withholding atezolizumab, permanently discontinue<br/>atezolizumab and contact Medical Monitor.</li> </ul> |
| or | |
| AST/ALT is >3×ULN to<br>≤5×ULN at baseline and<br>increases to<br>>8×ULN to ≤10×ULN | |
| AST or ALT increases to<br>>10×ULN or | Permanently discontinue atezolizumab and contact Medical<br>Monitor. O |
| total bilirubin increases to<br>> 3×ULN | <ul> <li>Consider patient referral to GI specialist for evaluation and<br/>liver biopsy to establish etiology of hepatic injury.</li> <li>Initiate treatment with corticosteroids equivalent to</li> </ul> |
| | 1–2 mg/kg/day oral prednisone. |
| | <ul> <li>If event does not improve within 48 hours after initiating<br/>corticosteroids, consider adding an immunosuppressive<br/>agent.</li> </ul> |
| | <ul> <li>If event resolves to baseline, taper corticosteroids over<br/>≥ 1 month.</li> </ul> |

GI=gastrointestinal; LFT=liver function test; ULN=upper limit of normal.

- a Atezolizumab may be withheld for a longer period of time (i.e., > 12 weeks after event onset) to allow for corticosteroids (if initiated) to be reduced to the equivalent of ≤ 10 mg/day oral prednisone. The acceptable length of the extended period of time must be based on assessment of benefit-risk by the investigator and in alignment with the protocol requirement for duration of treatment and documented by the investigator. Medical Monitor is available to advise as needed.
- If corticosteroids have been initiated, they must be tapered over ≥1 month to the equivalent of ≤10 mg/day oral prednisone before atezolizumab can be resumed.
- Resumption of atezolizumab may be considered in patients who are deriving benefit and have fully recovered from the immune-mediated event. The decision to rechallenge patients with atezolizumab should be based on investigator's assessment of benefit-risk and documented by the investigator (or an appropriate delegate). Medical Monitor is available to advise as needed.



#### **GASTROINTESTINAL EVENTS**

Immune-mediated colitis has been associated with the administration of atezolizumab. Management guidelines for diarrhea or colitis are provided in Table 3.

All events of diarrhea or colitis should be thoroughly evaluated for other more common etiologies. For events of significant duration or magnitude or associated with signs of systemic inflammation or acute-phase reactants (e.g., increased C-reactive protein, platelet count, or bandemia): Perform sigmoidoscopy (or colonoscopy, if appropriate) with colonic biopsy, with three to five specimens for standard paraffin block to check for inflammation and lymphocytic infiltrates to confirm colitis diagnosis.

**Table 3 Management Guidelines for Gastrointestinal Events (Diarrhea or Colitis)** 

| Event | Management |
|---|---|
| Diarrhea or colitis, Grade 1 | <ul> <li>Continue atezolizumab.</li> <li>Initiate symptomatic treatment.</li> <li>Endoscopy is recommended if symptoms persist for &gt;7 days.</li> <li>Monitor closely.</li> </ul> |
| Diarrhea or<br>colitis, Grade 2 | <ul> <li>Withhold atezolizumab for up to 12 weeks after event onset.<sup>3</sup></li> <li>Initiate symptomatic treatment.</li> <li>Patient referral to GI specialist is recommended.</li> <li>For recurrent events or events that persist &gt; 5 days, initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day oral prednisone.</li> <li>If event resolves to Grade 1 or better, resume atezolizumab.<sup>5</sup></li> <li>If event does not resolve to Grade 1 or better while withholding atezolizumab, permanently discontinue atezolizumab and contact Medical Monitor.<sup>5</sup></li> </ul> |
| Diarrhea or<br>colitis, Grade 3 | <ul> <li>Withhold atezolizumab for up to 12 weeks after event onset.<sup>a</sup></li> <li>Refer patient to GI specialist for evaluation and confirmatory biopsy.</li> <li>Initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day IV methylprednisolone and convert to 1–2 mg/kg/day oral prednisone or equivalent upon improvement.</li> <li>If event resolves to Grade 1 or better, resume atezolizumab.<sup>b</sup></li> <li>If event does not resolve to Grade 1 or better while withholding atezolizumab, permanently discontinue atezolizumab and contact Medical Monitor.<sup>c</sup></li> </ul> |



| Event | Management |
|---|---|
| Diarrhea or colitis, Grade 4 | <ul> <li>Permanently discontinue atezolizumab and contact Medical Monitor.</li> <li>Refer patient to GI specialist for evaluation and confirmatory biopsy.</li> <li>Initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day IV methylprednisolone and convert to 1–2 mg/kg/day oral prednisone or equivalent upon improvement.</li> <li>If event does not improve within 48 hours after initiating corticosteroids, consider adding an immunosuppressive agent.</li> <li>If event resolves to Grade 1 or better, taper corticosteroids over ≥1 month.</li> </ul> |

- a Atezolizumab may be withheld for a longer period of time (i.e., > 12 weeks after event onset) to allow for corticosteroids (if initiated) to be reduced to the equivalent of ≤ 10 mg/day oral prednisone. The acceptable length of the extended period of time must be based on assessment of benefit-risk by the investigator and in alignment with the protocol requirement for duration of treatment and documented by the investigator. Medical Monitor is available to advise as needed.
- b If corticosteroids have been initiated, they must be tapered over ≥1 month to the equivalent of ≤10 mg/day oral prednisone before atezolizumab can be resumed.
- Resumption of atezolizumab may be considered in patients who are deriving benefit and have fully recovered from the immune-mediated event. The decision to rechallenge patients with atezolizumab should be based on investigator's assessment of benefit-risk and documented by the investigator (or an appropriate delegate). Medical Monitor is available to advise as needed.

#### **ENDOCRINE EVENTS**

Thyroid disorders, adrenal insufficiency, diabetes mellitus, and pituitary disorders have been associated with the administration of atezolizumab. Management guidelines for endocrine events are provided in Table 4.

Patients with unexplained symptoms such as headache, fatigue, myalgias, impotence, constipation, or mental status changes should be investigated for the presence of thyroid, pituitary, or adrenal endocrinopathies. The patient should be referred to an endocrinologist if an endocrinopathy is suspected. Thyroid-stimulating hormone (TSH) and free triiodothyronine and thyroxine levels should be measured to determine whether thyroid abnormalities are present. Pituitary hormone levels and function tests (e.g., TSH, growth hormone, luteinizing hormone, follicle-stimulating hormone, testosterone, prolactin, adrenocorticotropic hormone [ACTH] levels, and ACTH stimulation test) and magnetic resonance imaging (MRI) of the brain (with detailed pituitary sections) may help to differentiate primary pituitary insufficiency from primary adrenal insufficiency.



# **Table 4 Management Guidelines for Endocrine Events**

| Event | Management |
|---|---|
| Asymptomatic<br>hypothyroidism | Continue atezolizumab. Initiate treatment with thyroid replacement hormone. Monitor TSH closely. |
| Symptomatic<br>hypothyroidism | Withhold atezolizumab. Initiate treatment with thyroid replacement hormone. Monitor TSH closely. Consider patient referral to endocrinologist. Resume atezolizumab when symptoms are controlled and thyroid function is improving. |
| Asymptomatic<br>hyperthyroidism | TSH≥0.1 mU/L and <0.5 mU/L: Continue atezolizumab. Monitor TSH every 4 weeks. Consider patient referral to endocrinologist. TSH <0.1 mU/L: Follow guidelines for symptomatic hyperthyroidism. Consider patient referral to endocrinologist. |
| Symptomatic<br>hyperthyroidism | <ul> <li>Withhold atezolizumab.</li> <li>Initiate treatment with anti-thyroid drug such as methimazole or carbimazole as needed.</li> <li>Consider patient referral to endocrinologist.</li> <li>Resume atezolizumab when symptoms are controlled and thyroid function is improving.</li> <li>Permanently discontinue atezolizumab and contact Medical Monitor for life-threatening immune-mediated hyperthyroidism.<sup>c</sup></li> </ul> |


| Event | Management |
|---|---|
| Symptomatic adrenal insufficiency, Grades 2–4 | Withhold atezolizumab for up to 12 weeks after event onset. Refer patient to endocrinologist. Perform appropriate imaging. |
| | <ul> <li>Initiate treatment with corticosteroids equivalent to<br/>1–2 mg/kg/day IV methylprednisolone and convert to<br/>1–2 mg/kg/day oral prednisone or equivalent upon<br/>improvement.</li> </ul> |
| | <ul> <li>If event resolves to Grade 1 or better and patient is stable on<br/>replacement therapy, resume atezolizumab.</li> </ul> |
| | <ul> <li>If event does not resolve to Grade 1 or better or patient is not<br/>stable on replacement therapy while withholding atezolizumab,<br/>permanently discontinue atezolizumab and contact Medical<br/>Monitor.<sup>c</sup></li> </ul> |
| Hyperglycemia,<br>Grade 1 or 2 | <ul> <li>Continue atezolizumab.</li> <li>Investigate for diabetes. If patient has Type 1 diabetes, treat as a Grade 3 event. If patient does not have Type 1 diabetes, treat as per institutional guidelines.</li> <li>Monitor for glucose control.</li> </ul> |
| Hyperglycemia,<br>Grade 3 or 4 | Withhold atezolizumab. Initiate treatment with insulin. Evaluate for diabetic ketoacidosis and manage as per institutional guidelines. Monitor for glucose control. Resume atezolizumab when symptoms resolve and glucose levels are stable. |



| Event | Management |
|---|---|
| Hypophysitis<br>(pan-hypopituitarism),<br>Grade 2 or 3 | <ul> <li>Withhold atezolizumab for up to 12 weeks after event onset.<sup>a</sup></li> <li>Refer patient to endocrinologist.</li> <li>Perform brain MRI (pituitary protocol).</li> <li>Initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day IV methylprednisolone and convert to 1–2 mg/kg/day oral prednisone or equivalent upon improvement.</li> <li>Initiate hormone replacement if clinically indicated.</li> <li>If event resolves to Grade 1 or better, resume atezolizumab.<sup>b</sup></li> <li>If event does not resolve to Grade 1 or better while withholding atezolizumab, permanently discontinue atezolizumab and contact Medical Monitor.<sup>c</sup></li> <li>For recurrent hypophysitis, treat as a Grade 4 event.</li> </ul> |
| Hypophysitis<br>(pan-hypopituitarism),<br>Grade 4 | Permanently discontinue atezolizumab and contact Medical Monitor. Refer patient to endocrinologist. Perform brain MRI (pituitary protocol). Initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day IV methylprednisolone and convert to 1–2 mg/kg/day oral prednisone or equivalent upon improvement. Initiate hormone replacement if clinically indicated. |

- <sup>a</sup> Atezolizumab may be withheld for a longer period of time (i.e., > 12 weeks after event onset) to allow for corticosteroids (if initiated) to be reduced to the equivalent of ≤ 10 mg/day oral prednisone. The acceptable length of the extended period of time must be based on assessment of benefit-risk by the investigator and in alignment with the protocol requirement for duration of treatment and documented by the investigator. Medical Monitor is available to advise as needed.
- b If corticosteroids have been initiated, they must be tapered over ≥1 month to the equivalent of ≤10 mg/day oral prednisone before atezolizumab can be resumed.
- Resumption of atezolizumab may be considered in patients who are deriving benefit and have fully recovered from the immune-mediated event. The decision to rechallenge patients with atezolizumab should be based on investigator's assessment of benefit-risk and documented by the investigator (or an appropriate delegate). Medical Monitor is available to advise as needed.

# **OCULAR EVENTS**

An ophthalmologist should evaluate visual complaints (e.g., uveitis, retinal events). Management guidelines for ocular events are provided in Table 5.



# **Table 5 Management Guidelines for Ocular Events**

| Event | Management |
|---|---|
| Ocular event,<br>Grade 1 | Continue atezolizumab. Patient referral to ophthalmologist is strongly recommended. Initiate treatment with topical corticosteroid eye drops and topical immunosuppressive therapy. |
| Ocular event,<br>Grade 2 | <ul> <li>Withhold atezolizumab for up to 12 weeks after event onset. <sup>a</sup></li> <li>Patient referral to ophthalmologist is strongly recommended.</li> <li>Initiate treatment with topical corticosteroid eye drops and topical immunosuppressive therapy.</li> <li>If event resolves to Grade 1 or better, resume atezolizumab. <sup>b</sup></li> <li>If event does not resolve to Grade 1 or better while withholding atezolizumab, permanently discontinue atezolizumab and contact Medical Monitor. <sup>c</sup></li> </ul> |
| Ocular event,<br>Grade 3 or 4 | <ul> <li>Permanently discontinue atezolizumab and contact Medical Monitor. <sup>c</sup></li> <li>Refer patient to ophthalmologist.</li> <li>Initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day oral prednisone.</li> <li>If event resolves to Grade 1 or better, taper corticosteroids over ≥1 month.</li> </ul> |

- <sup>a</sup> Atezolizumab may be withheld for a longer period of time (i.e., > 12 weeks after event onset) to allow for corticosteroids (if initiated) to be reduced to the equivalent of ≤10 mg/day oral prednisone. The acceptable length of the extended period of time must be based on assessment of benefit-risk by the investigator and in alignment with the protocol requirement for duration of treatment and documented by the investigator. Medical Monitor is available to advise as needed.
- b If corticosteroids have been initiated, they must be tapered over ≥1 month to the equivalent of ≤10 mg/day oral prednisone before atezolizumab can be resumed.
- Resumption of atezolizumab may be considered in patients who are deriving benefit and have fully recovered from the immune-mediated event. The decision to rechallenge patients with atezolizumab should be based on investigator's assessment of benefit-risk and documented by the investigator (or an appropriate delegate). Medical Monitor is available to advise as needed.

# **IMMUNE-MEDIATED MYOCARDITIS**

Immune-mediated myocarditis has been associated with the administration of atezolizumab. Immune-mediated myocarditis should be suspected in any patient presenting with signs or symptoms suggestive of myocarditis, including, but not limited to, laboratory (e.g., BNP [B-Natriuretic Peptide]) or cardiac imaging abnormalities, dyspnea, chest pain, palpitations, fatigue, decreased exercise tolerance, or syncope. Myocarditis may also be a clinical manifestation of myositis and should be managed accordingly Immune-mediated myocarditis needs to be



distinguished from myocarditis resulting from infection (commonly viral, e.g., in a patient who reports a recent history of gastrointestinal illness), ischemic events, underlying arrhythmias, exacerbation of preexisting cardiac conditions, or progression of malignancy.

All patients with possible myocarditis should be urgently evaluated by performing cardiac enzyme assessment, an ECG, a chest X-ray, an echocardiogram, and a cardiac MRI as appropriate per institutional guidelines. A cardiologist should be consulted. An endomyocardial biopsy may be considered to enable a definitive diagnosis and appropriate treatment, if clinically indicated.

Patients with signs and symptoms of myocarditis, in the absence of an identified alternate etiology, should be treated according to the guidelines in Table 6.

**Table 6 Management Guidelines for Immune-Related Myocarditis** 

| Event | Management |
|---|---|
| Immune-mediated<br>myocarditis, Grades | Permanently discontinue atezolizumab and contact Medical Monitor. |
| 2-4 | Refer patient to cardiologist. |
| | <ul> <li>Initiate treatment as per institutional guidelines and consider<br/>antiarrhythmic drugs, temporary pacemaker, ECMO, or VAD<br/>as appropriate.</li> </ul> |
| | <ul> <li>Initiate treatment with corticosteroids equivalent to<br/>1–2 mg/kg/day IV methylprednisolone and convert to<br/>1–2 mg/kg/day oral prednisone or equivalent upon<br/>improvement.</li> </ul> |
| | <ul> <li>If event does not improve within 48 hours after initiating<br/>corticosteroids, consider adding an immunosuppressive agent.</li> </ul> |
| | <ul> <li>If event resolves to Grade 1 or better, taper corticosteroids<br/>over≥1 month.</li> </ul> |

ECMO = extracorporeal membrane oxygenation; VAD = ventricular assist device.

a Resumption of atezolizumab may be considered in patients who are deriving benefit and have fully recovered from the immune-mediated event. The decision to rechallenge patients with atezolizumab should be based on investigator's assessment of benefit-risk and documented by the investigator (or an appropriate delegate). Medical Monitor is available to advise as needed.



#### INFUSION-RELATED REACTIONS AND CYTOKINE-RELEASE SYNDROME

No premedication is indicated for the administration of Cycle 1 of atezolizumab. However, patients who experience an infusion-related reaction (IRR) or cytokine-release syndrome (CRS) with atezolizumab may receive premedication with antihistamines, anti-pyretics, and/or analgesics (e.g., acetaminophen) for subsequent infusions. Metamizole (dipyrone) is prohibited in treating atezolizumab-associated IRRs because of its potential for causing agranulocytosis.

IRRs are known to occur with the administration of monoclonal antibodies and have been reported with atezolizumab. These reactions, which are thought to be due to release of cytokines and/or other chemical mediators, occur within 24 hours of atezolizumab administration and are generally mild to moderate in severity.

CRS is defined as a supraphysiologic response following administration of any immune therapy that results in activation or engagement of endogenous or infused T cells and/or other immune effector cells. Symptoms can be progressive, always include fever at the onset, and may include hypotension, capillary leak (hypoxia), and end-organ dysfunction (Lee et al. 2019). CRS has been well documented with chimeric antigen receptor T-cell therapies and bispecific T-cell engager antibody therapies but has also been reported with immunotherapies that target PD-1 or PD-L1 (Rotz et al. 2017; Adashek and Feldman 2019), including atezolizumab.

There may be significant overlap in signs and symptoms of IRRs and CRS, and in recognition of the challenges in clinically distinguishing between the two, consolidated guidelines for medical management of IRRs and CRS are provided in table 7.

Severe COVID-19 appears to be associated with a cytokine-release syndrome (CRS) involving the inflammatory cytokines interleukin (IL)-6, IL-10, IL-2, and interferon- $\gamma$  (Merad and Martin 2020). If a patient develops suspected CRS during the study, a differential diagnosis should include COVID-19, which should be confirmed or refuted through assessment of exposure history, appropriate laboratory testing, and clinical or radiologic evaluations per investigator judgment. If a diagnosis of COVID-19 is confirmed, the disease should be managed as per local or institutional guidelines.



# Table 7 Management Guidelines for Infusion-Related Reactions and Cytokine-Release Syndrome

| Event | Management |
|---|---|
| Grade 1 a fever b with or without constitutional symptoms | <ul> <li>Immediately interrupt infusion.</li> <li>Upon symptom resolution, wait for 30 minutes and then restart infusion at half the rate being given at the time of event onset.</li> <li>If the infusion is tolerated at the reduced rate for 30 minutes, the infusion rate may be increased to the original rate.</li> <li>If symptoms recur, discontinue infusion of this dose.</li> <li>Administer symptomatic treatment, or including maintenance of IV fluids for hydration.</li> <li>In case of rapid decline or prolonged CRS (&gt;2 days) or in patients with significant symptoms and/or comorbidities, consider managing as per Grade 2.</li> <li>For subsequent infusions, consider administration of oral premedication with antihistamines, anti-pyretics, and/or analgesics,</li> </ul> |
| Grade 23 | and monitor closely for IRRs and/or CRS. |
| Grade 2 a fever b with hypotension not requiring vasopressors and/or hypoxia requiring low-flow oxygen by nasal cannula or blow-by | <ul> <li>Immediately interrupt infusion.</li> <li>Upon symptom resolution, wait for 30 minutes and then restart infusion at half the rate being given at the time of event onset.</li> <li>If symptoms recur, discontinue infusion of this dose.</li> <li>Administer symptomatic treatment.<sup>c</sup></li> <li>For hypotension, administer IV fluid bolus as needed.</li> <li>Monitor cardiopulmonary and other organ function closely (in the ICU, if appropriate). Administer IV fluids as clinically indicated and manage constitutional symptoms and organ toxicities as per institutional practice.</li> <li>Rule out other inflammatory conditions that can mimic CRS (e.g., sepsis). If no improvement within 24 hours, initiate workup and assess for signs and symptoms of HLH or MAS.</li> <li>Consider IV corticosteroids (e.g., methylprednisolone 2 mg/kg/day or dexamethasone 10 mg every 6 hours).</li> <li>Consider anti-cytokine therapy.</li> <li>Consider hospitalization until complete resolution of symptoms. If no improvement within 24 hours, manage as per Grade 3, that is, hospitalize patient (monitoring in the ICU is recommended), permanently discontinue atezolizumab, and contact Medical</li> </ul> |
| | <ul> <li>Monitor.</li> <li>If symptoms resolve to Grade 1 or better for 3 consecutive days, next dose of atezolizumab may be administered. For subsequent infusions, consider administration of oral premedication with antihistamines, anti-pyretics, and/or analgesics and monitor closely for IRRs and/or CRS.</li> <li>If symptoms do not resolve to Grade 1 or better for 3 consecutive days, contact Medical Monitor.</li> </ul> |



| Event | Management |
|---|---|
| Grade 3ª fever® with hypotension requiring a vasopressor (with or without vasopressin) and/or hypoxia requiring high-flow oxygen® by nasal cannula, face mask, non-rebreather mask, or venturi mask | <ul> <li>Permanently discontinue atezolizumab and contact Medical Monitor. e</li> <li>Administer symptomatic treatment. c</li> <li>For hypotension, administer IV fluid bolus and vasopressor as needed.</li> <li>Monitor cardiopulmonary and other organ function closely; monitoring in the ICU is recommended. Administer IV fluids as clinically indicated, and manage constitutional symptoms and organ toxicities as per institutional practice.</li> <li>Rule out other inflammatory conditions that can mimic CRS (e.g., sepsis). If no improvement within 24 hours, initiate workup and assess for signs and symptoms of HLH or MAS.</li> <li>Administer IV corticosteroids (e.g., methylprednisolone 2 mg/kg/day or dexamethasone 10 mg every 6 hours).</li> <li>Consider anti-cytokine therapy.</li> <li>Hospitalize patient until complete resolution of symptoms. If no improvement within 24 hours, manage as per Grade 4, that is, admit patient to ICU and initiate hemodynamic monitoring, mechanical ventilation, and/or IV fluids and vasopressors as needed; for patients who are refractory to anti-cytokine therapy, experimental treatments may be considered at the discretion of the investigator and in consultation with the Medical Monitor.</li> </ul> |
| Grade 4 a fever b with hypotension requiring multiple vasopressors (excluding vasopressin) and/or hypoxia requiring oxygen by positive pressure (e.g., CPAP, BiPAP, intubation and mechanical ventilation) | <ul> <li>Permanently discontinue atezolizumab and contact Medical Monitor. <sup>e</sup></li> <li>Administer symptomatic treatment. <sup>e</sup></li> <li>Admit patient to ICU and initiate hemodynamic monitoring, mechanical ventilation, and/or IV fluids and vasopressors as needed. Monitor other organ function closely. Manage constitutional symptoms and organ toxicities as per institutional practice.</li> <li>Rule out other inflammatory conditions that can mimic CRS (e.g., sepsis). If no improvement within 24 hours, initiate workup and assess for signs and symptoms of HLH or MAS.</li> <li>Administer IV corticosteroids (e.g., methylprednisolone 2 mg/kg/day or dexamethasone 10 mg every 6 hours).</li> <li>Consider anti-cytokine therapy. For patients who are refractory to anti-cytokine therapy, experimental treatments<sup>r</sup> may be considered at the discretion of the investigator and in consultation with the Medical Monitor.</li> <li>Hospitalize patient until complete resolution of symptoms.</li> </ul> |



ASTCT=American Society for Transplantation and Cellular Therapy; BiPAP=bi-level positive airway pressure; CAR=chimeric antigen receptor; CPAP=continuous positive airway pressure; CRS=cytokine-release syndrome; CTCAE=Common Terminology Criteria for Adverse Events; eCRF=electronic Case Report Form; HLH=hemophagocytic lymphohistiocytosis; ICU=intensive care unit; IRR=infusion-related reaction; IV=intraveous; MAS=macrophage activation syndrome; NCCN=National Cancer Comprehensive Network; NCI=National Cancer Institute.

Note: These management guidelines have been adapted from the NCCN guidelines for the management of CAR T-cell-related toxicities (Version 2.2019).

- <sup>a</sup> Grading system for these management guidelines is based on ASTCT consensus grading for CRS. NCI CTCAE (version as specified in the protocol) should be used when reporting severity of IRRs, CRS, or organ toxicities associated with CRS on the Adverse Event eCRF. Organ toxicities associated with CRS should not influence overall CRS grading.
- <sup>b</sup> Fever is defined as temperature ≥38°C not attributable to any other cause. In patients who develop CRS and who then receive anti-pyretic, anti-cytokine, or corticosteroid therapy, fever is no longer required when subsequently determining event severity (grade). In this case, the grade is driven by the presence of hypotension and/or hypoxia.
- Symptomatic treatment may include oral or IV antihistamines, anti-pyretics, analgesics, bronchodilators, and/or oxygen. For bronchospasm, urticaria, or dyspnea, additional treatment may be administered as per institutional practice.
- d Low flow is defined as oxygen delivered at ≤ 6 L/min, and high flow is defined as oxygen delivered at > 6 L/min.
- Resumption of atezolizumab may be considered in patients who are deriving benefit and have fully recovered from the immune-mediated event. The decision to rechallenge patients with atezolizumab should be based on investigator's assessment of benefit-risk and documented by the investigator (or an appropriate delegate). Medical Monitor is available to advise as needed. For subsequent infusions, administer oral premedication with antihistamines, anti-pyretics, and/or analgesics, and monitor closely for IRRs and/or CRS. Premedication with corticosteroids and extending the infusion time may also be considered after assessing the benefit-risk ratio.
- <sup>1</sup> Refer to Riegler et al. (2019)

# PANCREATIC EVENTS

Symptoms of abdominal pain associated with elevations of amylase and lipase, suggestive of pancreatitis, have been associated with the administration of atezolizumab.

The differential diagnosis of acute abdominal pain should include pancreatitis. Appropriate workup should include an evaluation for ductal obstruction, as well as serum amylase and lipase tests. Management guidelines for pancreatic events, including pancreatitis, are provided in Table 8.



# Table 8 Management Guidelines for Pancreatic Events, Including Pancreatitis

| Event | Management |
|---|---|
| Amylase and/or lipase elevation, Grade 2 | Amylase and/or lipase > 1.5–2.0 × ULN: Continue atezolizumab. Monitor amylase and lipase weekly. For prolonged elevation (e.g., > 3 weeks), consider |
| | treatment with corticosteroids equivalent to 10 mg/day oral<br>prednisone. |
| | Asymptomatic with amylase and/or lipase > 2.0–5.0 × ULN: • Treat as Grade 3. |
| Amylase and/or lipase<br>elevation, Grade 3 or 4 | Withhold atezolizumab for up to 12 weeks after event onset. a |
| | Refer patient to GI specialist. |
| | <ul> <li>Monitor amylase and lipase every other day.</li> </ul> |
| | <ul> <li>If no improvement, consider treatment with corticosteroids<br/>equivalent to 1–2 mg/kg/day oral prednisone.</li> </ul> |
| | <ul> <li>If event resolves to Grade 1 or better, resume<br/>atezolizumab.</li> </ul> |
| | <ul> <li>If event does not resolve to Grade 1 or better while<br/>withholding atezolizumab, permanently discontinue<br/>atezolizumab and contact Medical Monitor.</li> </ul> |
| | <ul> <li>For recurrent events, permanently discontinue atezolizumab<br/>and contact Medical Monitor.</li> </ul> |



| Event | Management |
|---|---|
| Immune-mediated pancreatitis, Grade 2 or 3 | <ul> <li>Withhold atezolizumab for up to 12 weeks after event<br/>onset.<sup>a</sup></li> </ul> |
| | <ul> <li>Refer patient to GI specialist.</li> </ul> |
| | <ul> <li>Initiate treatment with corticosteroids equivalent to<br/>1–2 mg/kg/day IV methylprednisolone and convert to<br/>1–2 mg/kg/day oral prednisone or equivalent upon<br/>improvement.</li> </ul> |
| | <ul> <li>If event resolves to Grade 1 or better, resume<br/>atezolizumab.</li> </ul> |
| | <ul> <li>If event does not resolve to Grade 1 or better while<br/>withholding atezolizumab, permanently discontinue<br/>atezolizumab and contact Medical Monitor.</li> </ul> |
| | <ul> <li>For recurrent events, permanently discontinue atezolizumab<br/>and contact Medical Monitor.</li> </ul> |
| Immune-mediated pancreatitis, Grade 4 | Permanently discontinue atezolizumab and contact Medical<br>Monitor. One of the contact Medical Monitor. |
| | <ul> <li>Refer patient to GI specialist.</li> </ul> |
| | <ul> <li>Initiate treatment with corticosteroids equivalent to<br/>1–2 mg/kg/day IV methylprednisolone and convert to<br/>1–2 mg/kg/day oral prednisone or equivalent upon<br/>improvement.</li> </ul> |
| | <ul> <li>If event does not improve within 48 hours after initiating<br/>corticosteroids, consider adding an immunosuppressive<br/>agent.</li> </ul> |
| | <ul> <li>If event resolves to Grade 1 or better, taper corticosteroids<br/>over ≥ 1 month.</li> </ul> |

# GI=gastrointestinal.

- <sup>a</sup> Atezolizumab may be withheld for a longer period of time (i.e., > 12 weeks after event onset) to allow for corticosteroids (if initiated) to be reduced to the equivalent of ≤ 10 mg/day oral prednisone. The acceptable length of the extended period of time must be based on assessment of benefit-risk by the investigator and in alignment with the protocol requirement for duration of treatment and documented by the investigator. Medical Monitor is available to advise as needed.
- b If corticosteroids have been initiated, they must be tapered over ≥1 month to the equivalent of ≤10 mg/day oral prednisone before atezolizumab can be resumed.
- Resumption of atezolizumab may be considered in patients who are deriving benefit and have fully recovered from the immune-mediated event. The decision to rechallenge patients with atezolizumab should be based on investigator's assessment of benefit-risk and documented by the investigator (or an appropriate delegate). Medical Monitor is available to advise as needed.



## **DERMATOLOGIC EVENTS**

Treatment-emergent rash has been associated with atezolizumab. The majority of cases of rash were mild in severity and self limited, with or without pruritus. Although uncommon, cases of severe cutaneous adverse reactions such as Stevens-Johnson syndrome and toxic epidermal necrolysis have been reported with atezolizumab. A dermatologist should evaluate persistent and/or severe rash or pruritus. A biopsy should be considered unless contraindicated. Management guidelines for dermatologic events are provided in Table 9.

**Table 9 Management Guidelines for Dermatologic Events** 

| Event | Management |
|---|---|
| Dermatologic<br>event, Grade 1 | Continue atezolizumab. Consider treatment with topical corticosteroids and/or other symptomatic therapy (e.g., antihistamines). |
| Dermatologic<br>event, Grade 2 | <ul> <li>Continue atezolizumab.</li> <li>Consider patient referral to dermatologist for evaluation and, if indicated, biopsy.</li> <li>Initiate treatment with topical corticosteroids.</li> <li>Consider treatment with higher-potency topical corticosteroids if event does not improve.</li> <li>If unresponsive to topical corticosteroids, consider oral prednisone 0.5 mg/kg/day.</li> </ul> |
| Dermatologic<br>event, Grade 3 | <ul> <li>Withhold atezolizumab for up to 12 weeks after event onset.<sup>a</sup></li> <li>Refer patient to dermatologist for evaluation and, if indicated, biopsy.</li> <li>Initiate treatment with corticosteroids equivalent to 10 mg/day oral prednisone, increasing dose to 1–2 mg/kg/day if event does not improve within 48–72 hours.</li> <li>If event resolves to Grade 1 or better, resume atezolizumab.<sup>b</sup></li> <li>If event does not resolve to Grade 1 or better while withholding atezolizumab, permanently discontinue atezolizumab and contact Medical Monitor.<sup>c</sup></li> </ul> |
| Dermatologic<br>event, Grade 4 | Permanently discontinue atezolizumab and contact Medical Monitor. |
| Stevens-Johnson<br>syndrome or toxic<br>epidermal<br>necrolysis, (any<br>grade) | Additional guidance for Stevens-Johnson syndrome or toxic epidermal necrolysis: Withhold atezolizumab for suspected Stevens-Johnson syndrome or toxic epidermal necrolysis. Confirm diagnosis by referring patient to a specialist (dermatologist, ophthalmologist or urologist as relevant) for evaluation and, if indicated biopsy. Follow the applicable treatment and management guidelines above. If Stevens-Johnson syndrome or toxic epidermal necrolysis is confirmed, permanently discontinue atezolizumab. |



- a Atezolizumab may be withheld for a longer period of time (i.e., > 12 weeks after event onset) to allow for corticosteroids (if initiated) to be reduced to the equivalent of ≤10 mg/day oral prednisone. The acceptable length of the extended period of time must be based on assessment of benefit-risk by the investigator and in alignment with the protocol requirement for duration of treatment and documented by the investigator. Medical Monitor is available to advise as needed.
- If corticosteroids have been initiated, they must be tapered over ≥1 month to the equivalent of ≤10 mg/day oral prednisone before atezolizumab can be resumed.
- Resumption of atezolizumab may be considered in patients who are deriving benefit and have fully recovered from the immune-mediated event. The decision to rechallenge patients with atezolizumab should be based on investigator's assessment of benefit-risk and documented by the investigator (or an appropriate delegate). Medical Monitor is available to advise as needed.



#### **NEUROLOGIC DISORDERS**

Myasthenia gravis and Guillain-Barré syndrome have been observed with single-agent atezolizumab. Patients may present with signs and symptoms of sensory and/or motor neuropathy. Diagnostic work-up is essential for an accurate characterization to differentiate between alternative etiologies. Management guidelines for neurologic disorders are provided in Table 10.

**Table 10 Management Guidelines for Neurologic Disorders** 

| Event | Management |
|---|---|
| Immune-mediated<br>neuropathy, Grade<br>1 | Continue atezolizumab. Investigate etiology. |
| Immune-mediated<br>neuropathy, Grade<br>2 | Withhold atezolizumab for up to 12 weeks after event onset. Investigate etiology and refer patient to neurologist. Initiate treatment as per institutional guidelines. If event resolves to Grade 1 or better, resume atezolizumab. If event does not resolve to Grade 1 or better while withholding atezolizumab, permanently discontinue atezolizumab and contact Medical Monitor. Withhold atezolizumab for up to 12 weeks after event onset. In the second of the sec |
| Immune-mediated<br>neuropathy, Grade<br>3 or 4 | <ul> <li>Permanently discontinue atezolizumab and contact Medical Monitor.<sup>c</sup></li> <li>Refer patient to neurologist.</li> <li>Initiate treatment as per institutional guidelines.</li> </ul> |
| Myasthenia gravis<br>and Guillain-Barré<br>syndrome (any<br>grade) | <ul> <li>Permanently discontinue atezolizumab and contact Medical Monitor.<sup>c</sup></li> <li>Refer patient to neurologist.</li> <li>Initiate treatment as per institutional guidelines.</li> <li>Consider initiation of corticosteroids equivalent to 1–2 mg/kg/day oral or IV prednisone.</li> </ul> |

- a Atezolizumab may be withheld for a longer period of time (i.e., > 12 weeks after event onset) to allow for corticosteroids (if initiated) to be reduced to the equivalent of ≤ 10 mg/day oral prednisone. The acceptable length of the extended period of time must be based on assessment of benefit-risk by the investigator and in alignment with the protocol requirement for duration of treatment and documented by the investigator. Medical Monitor is available to advise as needed.
- If corticosteroids have been initiated, they must be tapered over ≥1 month to the equivalent of ≤10 mg/day oral prednisone before atezolizumab can be resumed.
- Resumption of atezolizumab may be considered in patients who are deriving benefit and have fully recovered from the immune-mediated event. The decision to rechallenge patients with atezolizumab should be based on investigator's assessment of benefit-risk and documented by the investigator (or an appropriate delegate). Medical Monitor is available to advise as needed.

# **IMMUNE-MEDIATED MENINGOENCEPHALITIS**

Immune-mediated meningoencephalitis is an identified risk associated with the administration of atezolizumab. Immune-mediated meningoencephalitis should be suspected in any patient



presenting with signs or symptoms suggestive of meningitis or encephalitis, including, but not limited to, headache, neck pain, confusion, seizure, motor or sensory dysfunction, and altered or depressed level of consciousness.

Encephalopathy from metabolic or electrolyte imbalances needs to be distinguished from potential meningoencephalitis resulting from infection (bacterial, viral, or fungal) or progression of malignancy, or secondary to a paraneoplastic process.

All patients being considered for meningoencephalitis should be urgently evaluated with a CT scan and/or MRI scan of the brain to evaluate for metastasis, inflammation, or edema. If deemed safe by the treating physician, a lumbar puncture should be performed and a neurologist should be consulted.

Patients with signs and symptoms of meningoencephalitis, in the absence of an identified alternate etiology, should be treated according to the guidelines in Table 11.

Table 11 Management Guidelines for Immune-Mediated Meningoencephalitis

| Event | Management |
|---|---|
| Immune-mediated<br>meningoencephalitis,<br>all grades | Permanently discontinue atezolizumab and contact Medical Monitor. <sup>a</sup> Refer patient to neurologist. |
| | <ul> <li>Initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day<br/>IV methylprednisolone and convert to 1–2 mg/kg/day oral<br/>prednisone or equivalent upon improvement.</li> </ul> |
| | <ul> <li>If event does not improve within 48 hours after initiating<br/>corticosteroids, consider adding an immunosuppressive agent.</li> </ul> |
| | <ul> <li>If event resolves to Grade 1 or better, taper corticosteroids over<br/>≥1 month.</li> </ul> |

<sup>&</sup>lt;sup>a</sup> Resumption of atezolizumab may be considered in patients who are deriving benefit and have fully recovered from the immune-mediated event. The decision to rechallenge patients with atezolizumab should be based on investigator's assessment of benefit-risk and documented by the investigator (or an appropriate delegate). Medical Monitor is available to advise as needed.

### **RENAL EVENTS**

Immune-mediated nephritis has been associated with the administration of atezolizumab. Eligible patients must have adequate renal function. Renal function, including serum creatinine, should be monitored throughout study treatment. Patients with abnormal renal function should be evaluated and treated for other more common etiologies (including prerenal and postrenal causes, and concomitant medications such as non-steroidal anti-inflammatory drugs). Refer the patient to a renal specialist if clinically indicated. A renal biopsy may be required to enable a definitive diagnosis and appropriate treatment.

Patients with signs and symptoms of nephritis, in the absence of an identified alternate etiology, should be treated according to the guidelines in Table 12.



**Table 12 Management Guidelines for Renal Events** 

| Event | Management |
|---|---|
| Renal event,<br>Grade 1 | <ul> <li>Continue atezolizumab.</li> <li>Monitor kidney function closely, including creatinine and urine protein<br/>until values resolve to within normal limits or to baseline values.</li> </ul> |
| Renal event,<br>Grade 2 | <ul> <li>Withhold atezolizumab for up to 12 weeks after event onset. <sup>a</sup></li> <li>Refer patient to renal specialist.</li> <li>Initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day oral prednisone.</li> <li>If event resolves to Grade 1 or better, resume atezolizumab. <sup>b</sup></li> <li>If event does not resolve to Grade 1 or better while withholding atezolizumab, permanently discontinue atezolizumab and contact Medical Monitor. <sup>c</sup></li> </ul> |
| Renal event,<br>Grade 3 or 4 | <ul> <li>Permanently discontinue atezolizumab and contact Medical Monitor.</li> <li>Refer patient to renal specialist and consider renal biopsy.</li> <li>Initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day oral prednisone.</li> <li>If event does not improve within 48 hours after initiating corticosteroids, consider adding an immunosuppressive agent.</li> <li>If event resolves to Grade 1 or better, taper corticosteroids over ≥ 1 month.</li> </ul> |

- a Atezolizumab may be withheld for a longer period of time (i.e., > 12 weeks after event onset) to allow for corticosteroids (if initiated) to be reduced to the equivalent of ≤ 10 mg/day oral prednisone. The acceptable length of the extended period of time must be based on assessment of benefit-risk by the investigator and in alignment with the protocol requirement for duration of treatment and documented by the investigator. Medical Monitor is available to advise as needed.
- b If corticosteroids have been initiated, they must be tapered over ≥1 month to the equivalent of ≤10 mg/day oral prednisone before atezolizumab can be resumed.
- Resumption of atezolizumab may be considered in patients who are deriving benefit and have fully recovered from the immune-mediated event. The decision to rechallenge patients with atezolizumab should be based on investigator's assessment of benefit-risk and documented by the investigator (or an appropriate delegate). Medical Monitor is available to advise as needed.

# **IMMUNE-MEDIATED MYOSITIS**

Myositis or inflammatory myopathies are a group of disorders sharing the common feature of inflammatory muscle injury; dermatomyositis and polymyositis are among the most common disorders. Initial diagnosis is based on clinical (muscle weakness, muscle pain, skin rash in dermatomyositis), biochemical (serum creatine kinase increase), and imaging (electromyography/MRI) features, and is confirmed with a muscle biopsy. Patients with possible myositis should be referred to a rheumatologist or neurologist. Patients with possible myositis should be monitored for signs of miocarditis.



Patients with signs and symptoms of myositis, in the absence of an identified alternate etiology, should be treated according to the guidelines in Table 13.

**Table 13 Management Guidelines for Immune-Mediated Myositis** 

| Event | Management |
|---|---|
| Immune-mediated<br>myositis, Grade 1 | Continue atezolizumab. Refer patient to rheumatologist or neurologist. Initiate treatment as per institutional guidelines. |
| Immune-mediated<br>myositis, Grade 2 | <ul> <li>Withhold atezolizumab for up to 12 weeks after event onset and contact Medical Monitor.</li> <li>Refer patient to rheumatologist or neurologist.</li> <li>Initiate treatment as per institutional guidelines.</li> <li>Consider treatment with corticosteroids equivalent to 1–2 mg/kg/day IV methylprednisolone and convert to 1–2 mg/kg/day oral prednisone or equivalent upon improvement.</li> <li>If corticosteroids are initiated and event does not improve within 48 hours after initiating corticosteroids, consider adding an immunosuppressive agent.</li> <li>If event resolves to Grade 1 or better, resume atezolizumab. b</li> <li>If event does not resolve to Grade 1 or better while withholding atezolizumab, permanently discontinue atezolizumab and contact Medical Monitor. c</li> </ul> |
| Immune-mediated myositis, Grade 3 | <ul> <li>Withhold atezolizumab for up to 12 weeks after event onset a and contact Medical Monitor.</li> <li>Refer patient to rheumatologist or neurologist.</li> <li>Initiate treatment as per institutional guidelines.</li> <li>Respiratory support may be required in more severe cases.</li> <li>Initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day IV methylprednisolone, or higher-dose bolus if patient is severely compromised (e.g., cardiac or respiratory symptoms, dysphagia, or weakness that severely limits mobility); convert to 1–2 mg/kg/day oral prednisone or equivalent upon improvement.</li> <li>If event does not improve within 48 hours after initiating corticosteroids consider adding an immunosuppressive agent.</li> <li>If event resolves to Grade 1 or better, resume atezolizumab. b</li> <li>If event does not resolve to Grade 1 or better while withholding atezolizumab, permanently discontinue atezolizumab and contact Medical Monitor.</li> <li>For recurrent events, treat as Grade 4 event. Permanently discontinue atezolizumab and contact Medical Monitor. c</li> </ul> |



| Event | Management |
|---|---|
| Immune-mediated<br>myositis, Grade 4 | <ul> <li>Permanently discontinue atezolizumab and contact Medical Monitor. °</li> <li>Refer patient to rheumatologist or neurologist.</li> <li>Initiate treatment as per institutional guidelines.</li> <li>Respiratory support may be required in more severe cases.</li> <li>Initiate treatment with corticosteroids equivalent to 1–2 mg/kg/day IV methylprednisolone, or higher-dose bolus if patient is severely compromised (e.g., cardiac or respiratory symptoms, dysphagia, or weakness that severely limits mobility); convert to 1–2 mg/kg/day oral prednisone or equivalent upon improvement.</li> </ul> |
| | <ul> <li>If event does not improve within 48 hours after initiating corticosteroids<br/>consider adding an immunosuppressive agent.</li> </ul> |
| | <ul> <li>If event resolves to Grade 1 or better, taper corticosteroids over<br/>≥1 month.</li> </ul> |

- a Atezolizumab may be withheld for a longer period of time (i.e., > 12 weeks after event onset) to allow for corticosteroids (if initiated) to be reduced to the equivalent of ≤ 10 mg/day oral prednisone. The acceptable length of the extended period of time must be based on assessment of benefit-risk by the investigator and in alignment with the protocol requirement for duration of treatment and documented by the investigator. Medical Monitor is available to advise as needed.
- b If corticosteroids have been initiated, they must be tapered over ≥1 month to the equivalent of ≤10 mg/day oral prednisone before atezolizumab can be resumed.
- Resumption of atezolizumab may be considered in patients who are deriving benefit and have fully recovered from the immune-mediated event. The decision to rechallenge patients with atezolizumab should be based on investigator's assessment of benefit-risk and documented by the investigator (or an appropriate delegate). Medical Monitor is available to advise as needed.

### HEMOPHAGOCYTIC LYMPHOHISTIOCYTOSIS AND MACROPHAGE ACTIVATION SYNDROME

Immune-mediated reactions may involve any organ system and may lead to hemophagocytic lymphohistiocytosis (HLH) and macrophage activation syndrome (MAS).

Clinical and laboratory features of severe CRS overlap with HLH, and HLH should be considered when CRS presentation is atypical or prolonged.

Patients with suspected HLH should be diagnosed according to published criteria by McClain and Eckstein (2014). A patient should be classified as having HLH if five of the following eight criteria are met:

Fever ≥ 38.5°C

Splenomegaly

Peripheral blood cytopenia consisting of at least two of the following:

- Hemoglobin < 90 g/L (9 g/dL) (< 100 g/L [10 g/dL] for infants < 4 weeks old)
- Platelet count  $< 100 \times 10^9 / L (100,000 / \mu L)$



- ANC  $< 1.0 \times 10^9 / L (1000 / \mu L)$ 

Fasting triglycerides > 2.992 mmol/L (265 mg/dL) and/or fibrinogen < 1.5 g/L (150 mg/dL) Hemophagocytosis in bone marrow, spleen, lymph node, or liver Low or absent natural killer cell activity

Ferritin > 500 mg/L (500 ng/mL)

Soluble IL-2 receptor (soluble CD25) elevated ≥ 2 standard deviations above age-adjusted laboratory-specific norms

Patients with suspected MAS should be diagnosed according to published criteria for systemic juvenile idiopathic arthritis by Ravelli et al. (2016). A febrile patient should be classified as having MAS if the following criteria are met:

Ferritin > 684 mg/L (684 ng/mL)

At least two of the following:

- − Platelet count ≤  $181 \times 10^9$ /L (181,000/μL)
- AST ≥ 48 U/L
- Triglycerides > 1.761 mmol/L (156 mg/dL)
- Fibrinogen  $\leq$  3.6 g/L (360 mg/dL)

Patients with suspected HLH or MAS should be treated according to the guidelines in Table 14.

Table 14 Management Guidelines for Suspected Hemophagocytic Lymphohistiocytosis or Macrophage Activation Syndrome

| Event | Management |
|---|---|
| Suspected HLH or MAS | <ul> <li>Permanently discontinue atezolizumab and contact Medical Monitor.</li> <li>Consider patient referral to hematologist.</li> <li>Initiate supportive care, including intensive care monitoring if indicated per institutional guidelines.</li> </ul> |
| | <ul> <li>Consider initiation of IV corticosteroids, an immunosuppressive agent,<br/>and/or anti-cytokine therapy.</li> </ul> |
| | <ul> <li>If event does not respond to treatment within 24 hours, contact Medical<br/>Monitor and initiate treatment as appropriate according to published<br/>guidelines (La Rosée 2015; Schram and Berliner 2015; La Rosée et al.<br/>2019).</li> </ul> |
| | <ul> <li>If event resolves to Grade 1 or better, taper corticosteroids over<br/>≥1 month.</li> </ul> |

HLH=hemophagocytic lymphohistiocytosis; IV=intravenous; MAS=macrophage activation syndrome.



# **APPENDIX 8**: Patient pre-screening form TELMA



Screening Form\_v.1.0\_11Apr2019

Av. Meridiana, 358 / 6ªplanta 08027 Barcelona Tel. 934 302 006 Fax. 934 191 766 Email: geop@geop.org www.geop.org

# TELMA (GECP 18/03-ML40237)

"A phase II open-label study of Atezolizumab in combination with bevacizumab as first line treatment for locally advanced or metastatic high-intermediate tumor mutation burden (TMB) selected non-squamous non-small cell lung cancer (NSCLC) patients"

## PRE-SCREENING FORM

Please send to Fundación GECP by Fax (Fax: 93 419 17 68) or

Email (Email: Imorales@gecp.org / asancho@gecp.org / averdu@gecp.org)

| PRE-SCREENING | NUMBER (A | ssigned by Fundación GEC | P) | |
|---|---|---|---|---|
| PRE-SCREENING | NUMBER: | st / / //_ | <del></del> | |
| | HOSPITA | AL DATA | | |
| HOSPITAL: | - | FAX OR EMAIL TO<br>RECEIVE RESULT: | | |
| INFORMED CO | NSENT, DAT | E OF BIRTH AND CRITERIA | į. | |
| INFORMED CONSENT DATE:// | <u> </u> | DATE OF BIRTH: | | X 8 |
| CRITERIA:<br>Does the patient comply with all incl | usion criteri | a and none of the exclusio | 500 | Yes<br>No |
| TUMOR SAMPLE:<br>Is there enough tumor sample for the | - | Yes<br>No<br>Unknown | | |
| SCREENING DATE:// | | NAME AND<br>SIGNATURE: | | |
| LABORATORY RES | ULTS (To be | filled out by Fundación Gl | ECP) | |
| SUFFICIENT SAMPLE: | □ Yes | □ No | □ NA | |
| TMB (≥10 mutations/ MB): | □ Yes | □ No | □ NA | |
| CAN THE PATIENT BE ENROLLED? | □ Yes | □ No, specify: | | |
| RESULTS DATE:// | | NAME AND<br>SIGNATURE: | | |

Protocol\_



# **APPENDIX 9:** Foundation one CDx Specimen Instructions



# Specimen Instructions

FoundationOne®CDx is an extensively validated tissue-based comprehensive genomic profiling service for all solid tumours. FoundationOne CDx analyses 324 cancer-related genes to provide potentially actionable information to help guide treatment options.1-3



# Acceptable Samples

- Formalin-fixed paraffin embedded (FFPE) specimens, including cut slide specimens are acceptable.
- Use standard fixation methods to preserve nucleic acid integrity. 10% neutral-buffered formalin for 6-72 hours is industry standard. DO NOT use other fixatives (Bouins, B5, AZF, Holland's).
- · Do not decalcify.

#### SAMPLE SIZE

When feasible, please send the block + 1 H&E slide.\*

10 unstained sildes (positively charged and unbaked at 4-5 microns thick) +1 H&E slide.\*





\*For smaller samples, providing the original H&E will preserve

### SURFACE AREA

MINIMUM: 25 mm<sup>2</sup>

If sending slides, provide 10 unstained slides cut at 4-5 microns thick to achieve a tissue volume of 1 mm<sup>1</sup>.\*\*



"Specimens with a smaller surface area may meet volume requirements by submitting additional unstained slides (USS) or block.

### TUMOUR CONTENT

OPTIMUM: 30% TN MINIMUM: 20% TN

Percent tumour nuclei (%TN) = number of tumour cells divided by total number of all cells with nuclei.

Note for liver specimens: higher tumour content may be required because hepatocyte nuclei have twice the DNA content of other somatic nuclei

## Shipping Instructions

- 1. Place the samples, FoundationOne CDx requisition form, and any other attachments into the FoundationOne CDx Specimen Shipping Kit.
- 2. Place the specimen shipping kit (including samples and paperwork) into the shipping pack, first ensuring that primary specimen containers (e.g. blocks, slides) are labelled with two patient-specific identifiers. Seal the shipping pack.
- 3. Complete the pre-printed shipping labels (If necessary) and apply to shipping pack.
- 4. Call to request a pick-up or drop the package at your site's designated pick-up location and ship sealed shipping pack to:

[insert local shipping information]

FoundationOne\*CDx is a next generation sequencing based in vitro diagnostic device for detection of substitutions, insertion and deletion alterations (indels) and copy number alterations (CNAs) in 324 genes and select gene rearrangements, as well as genomic signatures including turnour mutational burden (TMB) and microsatellite instability (MSI) using DNA isolated from formalin-fixed paraffin embodded (FFPE) turnour tissue specimens. The test is intended as a companion diagnostic to identify patients who may benefit from treatment with therapies in accordance with the approved therapeutic product labeling. Additionally, FoundationOne CDx is intended to provide turnour mutation profiling to be used by qualified health care professionals in accordance with professional guidelines in oncology for patients with solid malignant neoplasms.

For full information on the intended use, assay descriptions, and for detailed performance specifications, refer to the complete FoundationOne CDx label at rochefoundationmedicine.com

- 1. FoundationOne\*CDx FDA Approval, 2017. Available at: https://www.accessdata.fda.gov/cdrh.docs/pdf17/P170019a.pdf (Accessed August 2018)
  2. FoundationOne\*CDx FDA Approval Press Release, 2017. Available at: https://www.fda.gov/NewsEvents/Newsroom/PressAnnouncements/ucm5
- (Accessed August 2018).

  3. FoundationOne\*CDx Technical Specifications 2018. Available at: www.rochefoundationmedicine.com/ffcdxtech.

Foundation Medicine\* and FoundationOne\* are registered trademarks of Foundation Medicine\*, Inc. Roche is the licensed distributor of Foundation Medicine\* products outside of the United States [local affiliate contact details]

PR/FMI/1808/0015 Date of preparation: September 2018







# APPENDIX 10: Foundation one Liguid technical sheet

# **Technical Specifications**



FoundationOne\*Liquid is a liquid biopsy test for solid tumors that analyzes circulating tumor DNA (ctDNA) in blood.



### Clinical Background

Cell-free DNA (cfDNA) is DNA that circulates freely in the bloodstream. In a cancer patient, tumor cells that undergo apoptosis or necrosis also shed cell-free DNA. The tumor derived cell-free DNA is called circulating tumor DNA (ctDNA). By analyzing cell-free DNA isolated from a patient's blood, we can identify microsatellite instability (MSI)\* and clinically relevant genomic alterations in ctDNA and may match them to targeted therapies, immunotherapies and clinical trials.





#### Methods

FoundationOne Liquid:

- · Analyzes blood samples from patients with solid tumors including lung, breast, colon, etc.
- Uses a hybrid-capture, next-generation sequencing test method combined with proprietary computational algorithms that enable accurate variant calls by discriminating sequencing artifacts from bona fide mutations.
- Identifies four classes of genomic alterations (base substitutions, insertions and deletions, copy number alterations, and rearrangements), and reports high microsatellite instability.
- · Evaluates select clinically relevant genomic alterations in 70 commonly altered oncogenes.
- Features an optimized laboratory process to achieve high sensitivity and specificity, with enhanced extraction methodology to generate a large amount of high quality ctDNA.
- · Utilizes proprietary technology to accurately identify unique ctDNA fragments from plasma.

| | Mutant Allelle Frequency (MAF)/<br>Tumor Fraction <sup>1</sup> | Sensitivity <sup>2</sup> | Positive Predictive Value (PPV) |
|---|---|---|---|
| | > 0.5% | 99.9% (0.99.7% - 99.9%) | 100% (CI 99.9% - 100%) |
| Base substitutions | 0.25% - 0.5% | 95.8% (CI 94.5% - 96.9%) | 99.8% (C) 99.3% - 99.9%) |
| | 0.325% - 0.25% | % - 0.25% 68.4% (C) 65.7% - 70.9%) | |
| | > 0.5% | 99.7% (CI 98.7% - 99.9%) | 100% (CI 99.3% - 100%) |
| Insertions/Deletions<br>(Indels) (1-40bp) | 0.25% - 0.5% | 87.7% (CI 81.1% - 92.2%) | 98.8% (0 95.4% - 99.8%) |
| CONTRACTOR | 0.125% - 0.25% | 60.5% (Cr 52.7% - 67.7%) | 96.8% (CI 92.3% - 98.8%) |
| | > 0.5% | 700% (CI 85.9% - 100%) | 100% (CI 85.9% - 100%) |
| Rearrangements <sup>1</sup> | 0.25% - 0.5% | 89.4% (C) 65.5% - 96.2%) | 100% (CI 773% - 100%) |
| | 0.125% - 0.25% | 68.4% (CI 43.5% - 86.4%) | 100% (0171.7% - 100%) |
| Copy Number Amplifications | ≥ 20% | 95.3% (CI 82.9% - 99.2%). | 97.6% (CI 85.9% - 99.9%) |
| (CNA) <sup>4</sup> | < 20% | Varies depending on amplitude of<br>CNA and ctDNA fraction | |
| Microsatellite Instability (MSI) <sup>L</sup> | > 2.0% | 92.0% (C) 72.5% - 98.6%) | 100% (CI 82.2% -100%) |
| Reproducibility (average concordance between replicates) | | 97.7% Inter-batch precision<br>95.9% Intra-batch precision | |
| Specimen Type | | Peripheral whole blood (see Specimen Instructions for details) | |
| Turnaround Time <sup>6</sup> | | < 2 Weeks | |

Copy number amplifications were calculated using tumor fraction.
 95% confidence interval.
 Performance for gene fusions within targeted introns only. Sensitivity for gene fusions occurring outside targeted introns or in highly repetitive intronic sequence contexts is reduced.
 Copy number ≥ 8.
 Reported when MSI is determined to be high.
 Based on typical tumoround time from receipt of sample.





#### Reporting

- · Test results are provided in an interpretive report, curated by biomedical informatics scientists, and approved by board-certified and licensed pathologists.
- · Genomic findings are listed with clinically relevant targeted therapies, immunotherapies, and clinical trials.
- · Reported alterations may indicate response or lack of response to therapy (approved or in clinical trials), or may be drivers of oncogenesis based on reported scientific knowledge,
- · Reports include microsatellite instability (MSI)\* status, a biomarker that may help predict response to checkpoint inhibitors.
- Test results are available via our online portal at www.foundationmedicine.com<sup>†</sup> or by fax,

#### Additional Features

#### Mutant Allele Fraction (MAF)

The MAF listed denotes the frequency of the mutant allele identified in the sample. It is reported for base substitutions and insertions and deletions (indels).

#### Visualization of MAF

The clinical report includes a graphic representation of MAF. If multiple FoundationOne Liquid tests are ordered in the patient's treatment journey, the graphic will show the relative change in MAF which will allow treating physicians to better understand the evolution of a patient's disease and may help to inform the next steps in patient care.

#### Current Gene List<sup>‡</sup>

Entire coding sequence (base substitutions, indels, copy number alterations).

| | 3 4 | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| APC | AR | ATM | BRCAT | BRCA2 | CCND1 | CD274 (PD-L1) | CDH1 | CDK4 |
| CDK6 | CDK12 | CDKN2A | CHEK2 | CRKL. | EGFR | ERBB2 | ERRFIT | FGFR1 |
| FGFR2 | FOXL2 | KRAS | MDM2 | MET | MYC | MYCN | NFI | PALB2 |
| PDCD1LG2 | (PD-L2) | PTEN | PTPNII | RBI | SMO | STKII | TP53 | VEGFA |
| Select | Exons <sup>6</sup> | | | | | | | |
| ABLI | AKTI | ALK | ARAF | BRAF | BTK | CTNNB1 | DDR2 | ESR1 |
| EZH2 | FGFR3 | FLT3 | GNATI | GNAQ | GNAS | HRAS | IDHI | IDH2 |
| JAK2 | JAK3 | KIT | MAP2KT (MEKT) | MAP2K2 (MEK2) | MPL | MTOR | MYD88 | NPM1 |
| NRAS | PDGFRA | PDGFRB | PIK3CA | RAFI | RET | ROST | TERT | |
| Select | Rearrangeme | ents <sup>6</sup> | | | | | | |
| ALK | EGFR | FGFR2 | FGFR3 | PDGFRA | RET | ROS1 | | |

To learn more about our analytical validation based on a prior version of the test called FoundationACT (62 genes), see our publication in the Journal of Molecular Diagnostics: ""Analytical validation of a hybrid capture-based next-generation sequencing clinical assay for genomic profiling of cell-free circulating tumor DNA".

- Reported when MSI is determined to be high.
- Visit foundationmedicine.com to create an online account.

  Current as of August 2018. Please visit foundationmedicine.com for the most up-to-date gene list

F Detailed list available upon request.

Clark TA, et al. Analytical validation of a hybrid capture-based next-generation sequencing clinical assay for genomic profiling of cell-free circulating tumor DNA. J of Mol Diagn. 2018: published online ahead of print.



@ 2019 Foundation Medicine, Inc. | Foundation Medicine\* and FoundationOne\* are registered trademarks of Foundation Medicine, Inc. www.foundationmedicine.com | Tel. 888.988.3639 | Fax 617.418.2290 | MKT-0061-04

# **APPENDIX 11**: Foundation one CDx technical sheet

Please see documents attached to the protocol